## CLINICAL STUDY PROTOCOL

Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled,

Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of STS101 (Dihydroergotamine Nasal Powder) in the Acute Treatment of

Migraine

**Study Number:** STS101-007

**Investigational Drug:** STS101 (Dihydroergotamine Nasal Powder)

**IND Number:** 136585

**Sponsor:** Satsuma Pharmaceuticals, Inc.

400 Oyster Point Boulevard, Suite 221

South San Francisco, CA 94080

Tel. No.: 408-857-5248

Medical Monitor: Detlef Albrecht, MD

Tel. No.: 408-857-5248

**Version History:** Original March 8, 2021

Version 2 May 20, 2021

## **Confidentiality Statement**

The information contained in this document is the property of Satsuma Pharmaceuticals, Inc. and contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. In the event of any actual or suspected breach of this obligation, Satsuma Pharmaceuticals, Inc. should be promptly notified.

## **SIGNATURE PAGE (SPONSOR)**

I have read and understand the contents of this protocol and agree to meet all obligations of Satsuma Pharmaceuticals, Inc. as detailed in all applicable regulations and guidelines. In addition, I will ensure that the Principal Investigator is informed of all relevant information that becomes available during the conduct of the study.

Digitally signed by Detlef
Albrecht
Detlef Albrecht
Date:
2021.05.27
14:45:58 -07'00'

**Detlef Albrecht, MD**Chief Medical Officer
Satsuma Pharmaceuticals, Inc.

Date

## PRINCIPAL INVESTIGATOR AGREEMENT

I have carefully read this study protocol and agree that it contains all necessary information required to conduct this study. I agree to conduct the study according to this protocol (including any amendments) and in accordance with ICH Good Clinical Practices (GCP) and all other applicable regulations. I will inform all who assist me in the conduct of this study of their responsibilities and obligations. Furthermore, I understand that the Sponsor and the Institutional Review Board/Ethics Committee (IRB/EC) must approve any changes to the protocol in writing before implementation, unless a deviation is required to eliminate an immediate safety hazard to a subject. In such cases the Sponsor and the IRB/EC will be notified as soon as possible.

| Principal Investigator Signature | Date |
|-------------------------------------|------|
| Principal Investigator Name (print) | |
| Site Name | |

## PROTOCOL SYNOPSIS

| Sponsor/Company | Satsuma Pharmaceuticals, Inc. |
|---|---|
| Investigational<br>Product | STS101 (Dihydroergotamine Nasal Powder) |
| <b>Active Ingredient</b> | Dihydroergotamine mesylate |
| <b>Protocol Number</b> | STS101-007 |
| Title of Study | A Randomized, Double-Blind, Parallel Group, Placebo-Controlled,<br>Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of<br>STS101 (Dihydroergotamine Nasal Powder) in the Acute Treatment of<br>Migraine |
| Study center | Approximately 130 in the United States |
| <b>Objectives</b> | Primary |
| | <ul> <li>To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain at 2 hours after dosing</li> <li>To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve</li> </ul> |
| | freedom from most bothersome symptom at 2 hours after dosing |
| | Secondary |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid the use of rescue medication within 24 hours after dosing |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve normal function at 2 hours after dosing |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 24 hour sustained pain free status |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 48 hour sustained pain free status |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 24 hour sustained freedom from most bothersome symptom status |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 48 hour sustained freedom from most bothersome symptom status |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid the use of rescue medication within 48 hours after dosing |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid headache pain relapse within 24 hours after dosing |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid headache pain relapse within 48 hours after dosing |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain at various timepoints after dosing |
| | • To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from most bothersome symptom at various timepoints after dosing |

- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at various timepoints after dosing
- To estimate the probability of a subject to achieve freedom from pain during the 24-hour post dose period
- To estimate the probability of a subject to achieve freedom from the most bothersome symptom during the 24-hour post dose period
- To estimate the probability of a subject to achieve pain relief during the 24-hour post dose period
- To estimate the probability of a subject requiring rescue medication during the 24-hour post dose period
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from photophobia at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from phonophobia at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from nausea at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from photophobia at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from phonophobia at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from nausea at various timepoints after dosing
- To evaluate the study subject's global impression of the study treatment
- To assess the safety and tolerability of a single dose of 5.2 mg STS101 in the treatment of acute migraine attacks

#### **Exploratory**

- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain and most bothersome symptom by allodynia status at time of dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain and most bothersome symptom at 2 hours after dosing in subjects who wake up with acute migraine attacks
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain and most bothersome symptom at 2 hours after dosing in subjects with acute menstrual related migraine attacks
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing in subjects with acute migraine attacks by allodynia status at time of treatment
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing in subjects who wake up with acute migraine attacks

- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing in subjects with acute menstrual related migraine attacks
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve both, freedom from pain <u>and</u> most bothersome symptom at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve both, freedom from pain <u>and</u> most bothersome symptom at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from headache pain and most bothersome symptom (MBS) at 2 hours after dosing by baseline (Visit 2) HIT-6 score
- To evaluate the effects of a single dose of 5.2 mg STS101 on the 24-hour Migraine Quality of Life Questionnaire (24-MQoLQ)

## Methodology

This is a multi-center, single-dose, randomized, double-blind, placebo-controlled, parallel group study in approximately 1400 subjects with acute migraine (ages 18 to 65 years).

Study participants must have 2 to 8 migraine attacks, and fewer than 15 headache days during each of the three months before the screening visit.

At Visits 1 and 2, all study participants will be trained in the use of the STS101 device, the use of the electronic diary (e-diary) and undergo Placebo Response Reduction training, designed to improve discrimination between placebo and drug effects in clinical trials.

After establishing eligibility, the study participants will be randomized (1:1) to receive one of two treatments:

- 5.2 mg STS101 (equivalent to 6.0 mg of DHE mesylate USP)
- Placebo (matching nasal powder)

The randomization will be stratified by the use of migraine prevention medication. After the randomization, the study participants will treat their next qualifying migraine attack of at least moderate pain severity with the allocated blinded study medication within 4 hours of the onset of the attack.

The study participants will document the following symptoms of their treated migraine before and over 48 hours after study drug administration in an electronic diary (e-diary): migraine headache pain severity, presence of symptoms (photophobia, phonophobia, nausea), presence of allodynia and functionality status. Headache pain severity and symptom data will be documented immediately before drug administration (time 0), at 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after study drug administration. The subjects must select a most bothersome symptom among photophobia, phonophobia, and nausea immediately before study drug administration.

If subjects require rescue medication, they will be encouraged to wait until

the 2-hour post study drug administration data collection timepoint. The use of triptans or other DHE mesylate products as rescue medications should be avoided for 24 hours after study drug administration. The study participants will return to the study site within approximately one week of the treated migraine attack.

Adverse events, objective nasal evaluation data, safety laboratory data, vital sign data and ECGs will be recorded before and after treatment to evaluate the tolerability and safety of STS101.

# Number of subjects (planned)

A total of approximately 1400 adult male and female subjects aged 18 to 65 years with acute migraine headaches.

#### **Inclusion criteria**

- 1. English speaking males or females, 18-65 years of age at the time of Screening Visit
- 2. Signed Informed Consent Form
- 3. Subject has at least 1-year history of migraines (with or without aura), according to the International Classification of Headache Disorder, 3rd Edition (ICHD3), including the following:
  - a. Migraine onset before the age of 50 years
  - b. Migraine attacks, on average, lasting 4-72 hours if untreated
  - c. Migraine headache frequency of 2 to 8 attacks of moderate or severe pain intensity per month in each of the 3 months prior to the Screening Visit
  - d. Fewer than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit
  - e. Individual migraine attacks separated by at least 2 days of no headache pain
  - f. Subject is able to distinguish migraines from other headache types, e.g., tension-type or cluster headache.
- 4. Subjects on preventive migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to study entry and have no plans to change the dose during the study
- 5. Female subjects will be included if they are post-menopausal (at least 1 year since last menses with an FSH >40 IU/mL) or surgically sterilized; or if they are of childbearing potential, they are not breastfeeding, have a negative pregnancy test, have no intention of becoming pregnant during the course of the study, and are using one of the following medically acceptable contraceptive methods during the course of this study:
  - a. Simultaneous use of male condom and intra-uterine contraceptive device placed at least 4 weeks prior to screening (Visit 1)
  - b. Simultaneous use of male condom with intravaginally applied spermicide and diaphragm

- c. Simultaneous use of male condom and hormonal contraceptives started at least 4 weeks prior to screening (Visit 1)
- d. Surgical sterilization of their partner(s) at least 6 months prior to screening (Visit 1)
- 6. Intact nasal mucosa (Appendix C, Objective Assessment of Nasal Symptoms: no ulceration; no bleeding; no or mild erythema, no or mild swelling and no or mild rhinorrhea), and no other nasal conditions that may interfere with intranasal dosing at randomization (Visit 2)
- 7. Willing and able to comply with the requirements of the protocol and follow directions from the clinic staff
- 8. Adequate compliance (≥80%) in the completion of the e-diary during the Screening Period

#### Exclusion criteria

- 1. Pregnant or breast-feeding women
- 2. Women of child-bearing potential not using or not willing to use highly effective contraception
- 3. Diagnosis of headache conditions other than migraine with or without aura, including diagnosis of basilar or hemiplegic migraines, medication overuse headache or cluster headache
- 4. Abnormal physical findings of clinical significance which would interfere with the objectives of the study at the screening or randomization visit examination
- 5. History of coronary artery disease, coronary artery vasospasm (including Printz-metals' angina), clinically significant arrhythmia or, peripheral vascular disease, ischemic disease (e.g., Raynaud's syndrome, ischemic bowel syndrome, angina pectoris, myocardial infarction, or documented silent ischemia); percutaneous coronary intervention, or cardiac surgery
- 6. History of cerebrovascular disease, including but not limited to stroke, transient ischemic attack, cerebral hemorrhage, subarachnoid hemorrhage
- 7. Presence of two or more of the following cardiovascular risk factors:
  - a. Previous diagnosis of hypertension or currently taking antihypertensive medication
  - b. Previous diagnosis of hypercholesteremia, or currently taking cholesterol lowering treatment or LDL >159 mg/dL at screening (Visit 1; note: re-draws prior to Visit 2 may be permitted)
  - c. Obesity (BMI > 31)
  - d. Diabetes mellitus
  - e. Family history of premature coronary artery disease (in male first-degree relatives < 55 years or female first-degree relatives < 65 years)
  - f. Females who are surgically or physiologically postmenopausal

- g. Males 46 years and older
- 8. Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening (Visit 1; note: re-draws prior to Visit 2 may be permitted)
- 9. Severely impaired hepatic function (liver function tests ALT or AST greater than 2 times upper limit of normal) or renal function (serum creatinine greater than 1.5 times the upper limit of normal) at screening (Visit 1; note: re-draws prior to Visit 2 may be permitted)
- 10. Screening 12-lead ECG showing any clinically significant abnormalities at screening (Visit 1)
- 11. Systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, at screening (Visit 1)
- 12. Diagnosis of major depression with current symptoms, psychosis, alcohol abuse or dependence, drug abuse or dependence, major psychiatric conditions (e.g., schizophrenia, psychosis or Bipolar disorder), or dementia. Other significant neurological or psychiatric disorders (including other pain syndromes or risk of suicide) that in the opinion of the investigator might interfere with study participation and assessments or subject safety
- 13. Any clinically significant symptoms or conditions, including but not limited to central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator might interfere with study assessments or subject safety
- 14. Participation in another drug research study within 30 days of Screening Visit or within less than 5 half-lives of tested drug (whichever is longer)
- 15. Concomitant use of potent CYP3A4 inhibiting medications, for example protease inhibitors (e.g., ritonavir, nelfinavir, indinavir, saquinavir, tipranavir, lopinavir, atazanavir, darunavir), macrolide antibiotics (e.g., erythromycin, clarithromycin, troleandomycin), or strong imidazole antifungals (e.g., ketoconazole, and itraconazole)
- 16. Previously shown hypersensitivity to ergot alkaloids or the inactive ingredients of STS101 (microcrystalline cellulose, hydroxypropyl methylcellulose, mannitol)
- 17. Concomitant use of more than one preventive migraine medication.
- 18. Current use of opioids, cannabis or cannabinoid containing products
- 19. Concomitant use of peripheral and central vasoconstrictors including but not limited to amphetamines, phenylephrine, pseudoephedrine, propranolol and nicotine (from smoking, vaping or smokeless products)
- 20. Score of >0 on any of the questions 1-14 of the Sheehan Suicidality Tracking Scale

| <ul> <li>Investigational product, dosage and mode of administration</li> <li>5.2 mg STS101 dose strength (equivalent to 6.0 mg of DH USP; nasal powder)</li> <li>Placebo (matching nasal powder)</li> <li>For subject training</li> <li>STS101 Empty Training Devices</li> </ul> | |
|---|---|
| <b>Duration of study</b> | <ul> <li>STS101 Filled Training Devices (microcrystalline cellulose powder)</li> <li>Screening period: Up to 30 days</li> </ul> |
| • Treatment & follow up period: Up to 66 days | |
| Criteria for | Efficacy |
| Evaluation | Primary Efficacy: |
| | • Proportion of subjects free from headache pain at 2 hours after dosing (defined as moderate or severe headache pain [2 or 3 on a 4-point scale] at baseline [time 0] becoming none [0] on a 4-point scale) |
| | • Proportion of subjects free from most bothersome symptom (MBS) among photophobia, phonophobia and nausea at 2 hours after dosing (defined as the MBS selected at baseline [time 0] being absent) |
| | Secondary Efficacy: |
| | • Proportion of subjects with relief from headache pain at 2 hours after dosing (defined as reduction in headache pain from moderate or severe [2 or 3 on a 4-point scale] to mild or none [0 or 1 on a 4-point scale]) |
| | • Proportion of subjects who use rescue medication within 24 hours after dosing |
| | • Proportion of subjects who achieve normal function at 2 hours after dosing (defined as score of 0 on the 4-point functional impairment scale) |
| | • Proportion of subjects free from headache pain at 2 hours after dosing and remaining headache free at 24 hours after dosing with no use of rescue medication and no relapse of any headache pain (defined as score of 0 on a 4-point scale from 2-24 hours) |
| | • Proportion of subjects free from headache pain at 2 hours after dosing and remaining headache free at 48 hours after dosing with no use of rescue medication and no relapse of any headache pain (defined as score of 0 on a 4-point scale from 2-48 hours) |
| | • Proportion of subjects free from most bothersome symptom (MBS) at 2 hours after dosing and remaining MBS free at 24 hours after dosing with no use of rescue medication and no relapse of any MBS (defined as MBS selected at baseline [time 0] absent from 2-24 hours) |
| | • Proportion of subjects free from most bothersome symptom (MBS) at 2 hours after dosing and remaining MBS free at 48 hours after dosing with no use of rescue medication and no relapse of any MBS (defined as MBS selected at baseline [time 0] absent from 2-48 hours) |

- Proportion of subjects who use rescue medication within 48 hours after dosing
- Proportion of subjects with headache relapse within 24 hours after dosing (defined as the return of headache of any severity within 24 hours post dosing of the investigational drug, when the subject was pain-free at 2 hours after dosing)
- Proportion of subjects with headache relapse within 48 hours after dosing (defined as the return of headache of any severity within 48 hours post dosing of the investigational drug, when the subject was pain-free at 2 hours after dosing)
- Proportion of subjects free from headache pain at various time points after dosing
- Proportion of subjects free from most bothersome symptom at various time points after dosing
- Proportion of subjects achieving pain relief at various time points after dosing
- Proportion of subjects who achieve normal function at various timepoints after dosing
- Proportion of subjects free from photophobia (defined as photophobia being absent at 2 hours after dosing if present at baseline [time 0])
- Proportion of subjects free from phonophobia (defined as phonophobia being absent at 2 hours after dosing if present at baseline [time 0])
- Proportion of subjects free from nausea (defined as nausea being absent at 2 hours after dosing if present at baseline [time 0])
- Proportion of subjects free from photophobia at various timepoints after dosing
- Proportion of subjects free from phonophobia at various timepoints after dosing
- Proportion of subjects free from nausea at various timepoints after dosing
- Patient Global Impression ratings

## **Exploratory**

- Proportion of subjects free from headache pain at 2 hours after dosing by allodynia status at baseline (allodynia status will be defined as "present" with at least 2 "yes" responses to the 6-question allodynia questionnaire [Ashkenazi 2007; Tepper 2011])
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at 2 hours after dosing in subjects who wake up with migraine headache
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at 2 hours after dosing in subjects with menstrual related migraine attack

- Proportion of subjects with relief from headache pain at various timepoints after dosing by allodynia status at baseline (time 0) (allodynia status will be defined as "present" with at least 2 "yes" responses to the 6-question allodynia questionnaire [Ashkenazi 2007; Tepper 2011])
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at various timepoints after dosing in subjects who wake up with migraine headache
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at various timepoints after dosing in subjects with menstrual related migraine attack
- Proportion of subjects free from both, headache pain and most bothersome symptom (MBS) at 2 hours after dosing
- Proportion of subjects free from both, headache pain and most bothersome symptom (MBS) at various time points after dosing
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at 2 hours after dosing by baseline (Visit 2) HIT-6 score
- 24-hour Migraine Quality of Life Questionnaire summary scores

#### Safety

The following assessment and measurements will be conducted at screening, before randomization and at the final visit:

- Physical examination
- Vitals signs and body weight
- Objective nasal symptom assessment
- 12-lead ECG
- Blood tests for hematology and biochemistry analysis (including liver function, renal function, thyroid function, electrolytes)
- Urinalysis
- Adverse events (AEs)
- Documentation of concomitant medications

#### Statistical methods | Sample Size Determination

A total of approximately 1400 evaluable subjects is planned for the study. Given the 1:1 randomization ratio, approximately 700 subjects will be randomized to each treatment group. For the co-primary endpoint of pain freedom at 2 hours post dosing of investigational drug, a therapeutic gain of 10%, assuming a 25% responder rate for STS101 and 15% for the placebo is targeted. Based on these assumptions, 700 subjects per treatment group can provide 99% power to detect the target treatment difference. For the co-primary endpoint of MBS freedom at 2 hours post investigational drug, a therapeutic gain of 10%, assuming a 45% responder rate for STS101 and 35% for the placebo is targeted. Based on these assumptions, 700 subjects per treatment group can provide 95% power to detect the target treatment difference. The sample size calculation is based on a chi-square test with a significance level of 0.05 and a 2-sided test.

The primary efficacy objective will be addressed by simultaneously testing the 2 co-primary endpoints of pain freedom and MBS freedom at 2 hours after drug administration at a significance level of 0.05. This sample size will provide an overall power of at least 94%.

#### **Efficacy**

A detailed Statistical Analysis Plan (SAP) including the final hierarchy of testing of primary and secondary endpoints will be created before data base lock and study unblinding.

All study data will be summarized by treatment using descriptive statistics. Unless otherwise specified, for numeric data (e.g., age, weight), descriptive statistics will include the number of subjects with data to be summarized (n), mean, standard deviation (SD), median, minimum (min) and maximum (max). All categorical/qualitative data (e.g., gender, race) will be presented using absolute and relative frequency counts and percentage.

Data from all investigational centers will be pooled for analysis. For the primary analysis of the co-primary endpoints, missing data will be imputed based on a single-imputation method. Subjects who do not have evaluable assessments at the 2-hour time point, or who received rescue medications prior to the 2-hour time point will be considered as non-responders. The impact of missing data will be further investigated in a number of sensitivity analyses with other single and multiple-imputation approaches.

A study-wise Type I error of 0.05 will be used for this study. A fixed-sequence testing method with a pre-defined hierarchical order will be employed to control for the study-wise Type I error rate.

For both co-primary endpoints, the Chi-square test will be used to compare the active treatment groups and placebo. Chi-square test will also be used to test secondary endpoints consisting of proportion of responders. For analyses stratified by allodynia status, timing of treatment, the Cochran-Mantel-Haenszel test will be used. The Kaplan-Meier method will be used for time to use of rescue medications. The 24-hour Migraine Quality of Life Questionnaire assessments will be analyzed with the Analysis of Variance (ANOVA) models. The Chi-Square test will be used to analyze the Patient Global Impression ratings.

Subgroup analyses of the key efficacy endpoints will be conducted to gain insight of the nature and consistency of the treatment effect.

#### Safety

Safety analyses will include all subjects who received at least one dose of study medication.

All adverse events reported or observed will be listed, documenting severity, start and stop date and time, possible relationship to study medication, action taken, and outcome. Treatment emergent adverse events (TEAE) are defined as adverse events recorded after dosing of the investigational product. Verbatim terms will be classified to preferred terms (PT) and related system organ class (SOC) using the MedDRA dictionary. The preferred terms and system organ classes will be tabulated by treatment group. All reported adverse events will be summarized by the number of subjects reporting adverse events, system organ class, preferred term, severity and relationship to study drug.

Safety labs including complete blood count (CBC), chemistry and urinalysis will be tabulated using descriptive statistics. A tabulation of by-subject abnormal/out-of-range findings and changes from pre-dose (Visit 1) to post-dose in all laboratory variables will be provided.

Vital signs, objective and subjective evaluations of nasal symptom and standard 12-lead ECGs will be tabulated using descriptive statistics. A tabulation of by-subject abnormal/out-of-range findings and changes from pre-dose (Visit 1) to post-dose variables will be provided.

## **TABLE OF CONTENTS**

| Sig | nature | Page ( | Sponsor) | 2 |
|---|---|---|---|---|
| Pri | ncipal | Investi | gator Agreement | 3 |
| Pro | tocol | Synops | 18 | 4 |
| Lis | t of Ta | ables | | 19 |
| Lis | t of Fi | gures | | 19 |
| Lis | t of A | ppendic | ees | 19 |
| Lis | t of A | bbrevia | tions and Definitions of Terms | 20 |
| Stu | dy Pro | otocol F | Revision History | 22 |
| 1. | BAC | KGRO | UND INFORMATION | 24 |
| | 1.1. | Introd | uction | 24 |
| | 1.2. | STS10 | 01 Description | 25 |
| | | 1.2.1. | STS101 Device | 25 |
| | | 1.2.2. | STS101 Powder Formulation | 26 |
| | | | 1.2.2.1. DHE Mesylate Information | 26 |
| | | 1.2.3. | DHE Mechanism of Action in the Treatment of Migraine | 26 |
| | | 1.2.4. | STS101 DHE Pharmacokinetics | 26 |
| | | 1.2.5. | DHE Clinical Experience | 28 |
| | | 1.2.6. | DHE Mesylate Pregnancy Category | 28 |
| | 1.3. | Summ | nary of Nonclinical Data | 28 |
| | 1.4. | Summ | nary of Clinical Data for STS101 | 28 |
| | 1.5. | Ration | nale for the study | 29 |
| 2. | STU | DY OB | JECTIVES AND PURPOSE | 30 |
| 3. | STU | DY DE | SIGN | 32 |
| | 3.1. | Overa | ll Study Design and Plan | 32 |
| | 3.2. | Study | Procedures Descriptions | 33 |
| | | 3.2.1. | Informed Consent | 33 |
| | | 3.2.2. | Assignment of Subject Identification Number | 33 |
| | | 3.2.3. | Inclusion and Exclusion Criteria Assessment | 33 |
| | | 3.2.4. | Medical History, Demographics, Concomitant and Prior Medications | 33 |
| | | 3.2.5. | Headache Impact Test (HIT-6 <sup>TM</sup> ) | 34 |
| | | 3.2.6. | Physical Examination | 34 |
| | | 3.2.7. | Vital Signs | 34 |

| | | 3.2.8. | Weight, Height and Body Mass Index (BMI) | 34 |
|---|---|---|---|---|
| | | 3.2.9. | Evaluations of Effects in the Nose | 35 |
| | | | 3.2.9.1. Objective Assessment of Nasal Symptoms | 35 |
| | | 3.2.10 | . Clinical Laboratory Tests | 35 |
| | | | 3.2.10.1. Lab Testing for Chest Related Symptoms or Adverse Events | 36 |
| | | 3.2.11. | . Electrocardiogram | 36 |
| | | 3.2.12. | . Adverse Events Recording | 37 |
| | | 3.2.13 | . Electronic Headache Diary | 37 |
| | | 3.2.14. | . Placebo Response Reduction Training | 37 |
| | | 3.2.15. | . Sheehan Suicidality Tracking Scale (S-STS) | 37 |
| | 3.3. | Schedu | ule of Observations and Procedures | 37 |
| | | | Screening Procedures | |
| | | 3.3.2. | Screening Visit & Period (Day-30 to Day -1) | 38 |
| | | 3.3.3. | Randomization Visit (Visit 2; Day1) | 38 |
| | | 3.3.4. | Final Visit/Early Termination (Visit 3) | 39 |
| 4. | SELI | | N AND WITHDRAWAL OF SUBJECTS | |
| | 4.1. | Subjec | et Inclusion Criteria | 40 |
| | 4.2. | Subjec | et Exclusion Criteria | 41 |
| | 4.3. | Subjec | et Withdrawal Criteria | 42 |
| 5. | TRE | ATME | NT OF SUBJECTS | 44 |
| | 5.1. | Descri | ption of Investigational Product and Packaging | 44 |
| | 5.2. | Investi | igational Product Labeling | 44 |
| | 5.3. | Investi | igational Product Storage | 45 |
| | 5.4. | Investi | igational Product Administration & Training | 45 |
| | 5.5. | Investi | igational Product Accountability | 45 |
| | 5.6. | Investi | igational Product Handling and Disposal | 46 |
| | 5.7. | Conco | mitant Medications & Migraine Treatments | 46 |
| | 5.8. | Treatm | nent Compliance | 47 |
| | 5.9. | | mization and Blinding | |
| | | 5.9.1. | Subject Randomization | 47 |
| | | 5.9.2. | • | |
| | | 5.9.3. | Unblinding Procedures | |
| 6. | ASS | ESSME | NT OF EFFICACY | 48 |

| | 6.1. | Effica | cy Evaluation Parameters (e-Diary) | . 48 |
|---|---|---|---|---|
| | | 6.1.1. | Migraine Headache Pain Severity | . 48 |
| | | 6.1.2. | Most Bothersome Symptom | . 48 |
| | | 6.1.3. | Evaluation of Allodynia | . 48 |
| | | 6.1.4. | Use of Rescue Medication. | . 49 |
| | | 6.1.5. | Evaluation of Function | . 49 |
| | | | 6.1.5.1. Functional Impairment Scale | . 49 |
| | | | 6.1.5.2. 24-hour Migraine Quality of Life Questionnaire | . 49 |
| | 6.2. | Patien | t Subjective Impression Questions (Office; Visit 3) | . 50 |
| | | 6.2.1. | Patient Global Impression | . 50 |
| | | 6.2.2. | Ease of Use Impression | . 50 |
| | | 6.2.3. | Patient Likelihood of Use. | . 50 |
| | | 6.2.4. | Comparison of study medication with previously used migraine medication | . 50 |
| 7. | ASS | ESSME | NT OF SAFETY | 51 |
| | 7.1. | Safety | Parameters | . 51 |
| | | 7.1.1. | Examinations | . 51 |
| | | | 7.1.1.1. Physical Examinations | 51 |
| | | | 7.1.1.2. Height, Weight, and BMI | . 51 |
| | | | 7.1.1.3. Vital Signs | . 51 |
| | | | 7.1.1.4. Objective Nasal Symptom Assessments | 51 |
| | | | 7.1.1.5. Electrocardiogram (ECG) | . 51 |
| | | 7.1.2. | Laboratory Assessments | . 52 |
| | | | 7.1.2.1. Hematology | 52 |
| | | | 7.1.2.2. Serum Chemistry | . 52 |
| | | | 7.1.2.3. Urinalysis | . 52 |
| | | | 7.1.2.4. Urine Drug Screen | . 52 |
| | | | 7.1.2.5. Serum & Urine Pregnancy Test | . 52 |
| | | | 7.1.2.6. Serum FSH test | 52 |
| | | | 7.1.2.7. Lab testing for chest related symptoms or adverse events | 52 |
| | | | 7.1.2.8. Sheehan Suicidality Tracking Scale | . 53 |
| | 7.2. | Advers | se Events | . 53 |
| | | 7.2.1. | AE Relationship to Study Drug. | . 54 |
| | | 7.2.2. | Assessment of Adverse Event Severity | . 54 |

| | | 7.2.3. | Serious Adverse Events (SAEs) Recording and Reporting | 54 |
|---|---|---|---|---|
| 8. | STA | STATISTICS57 | | |
| | 8.1. | Sampl | le Size Determination | 57 |
| | 8.2. | Subjec | ct Populations | 57 |
| | | 8.2.1 | Intent-to-Treat Population | 57 |
| | | 8.2.2 | Modified Intent-to-Treat Population | 57 |
| | | 8.2.3 | Per-Protocol Population | 57 |
| | | 8.2.1. | Safety Population | 58 |
| | 8.3. | Statist | tical Analysis | 58 |
| | | 8.3.1. | Demographic and Baseline Variables | 58 |
| | | 8.3.2. | Efficacy Analysis | 58 |
| | | | 8.3.2.1. Primary Efficacy Endpoints | 58 |
| | | | 8.3.2.2. Secondary Efficacy Endpoints | 58 |
| | | | 8.3.2.3. Exploratory Endpoints | 59 |
| | | 8.3.3. | Hypotheses Testing and Significance Level | 60 |
| | | 8.3.4. | Handling of Missing Data | 60 |
| | | 8.3.5. | Pooling of Centers | 60 |
| | | 8.3.6. | Analysis Methods for Efficacy Endpoints | 61 |
| | | 8.3.7. | Subgroup Analysis of Efficacy Endpoints | 61 |
| | | 8.3.8. | Safety Analysis | 61 |
| | | | 8.3.8.1. Extent of Exposure | 62 |
| | | | 8.3.8.2. Adverse Events | 62 |
| | | | 8.3.8.3. Assessment of Nasal Symptoms | 62 |
| | | | 8.3.8.4. Laboratory Evaluations | 62 |
| | | | 8.3.8.5. Vital Signs | 63 |
| | | | 8.3.8.6. ECG Evaluations | 63 |
| | | | 8.3.8.7. Concomitant Medications | 63 |
| | | | 8.3.8.8. Sheehan Suicidality Tracking Scale | 63 |
| | | 8.3.9. | Interim analysis | 63 |
| 9. | DAT | 'A HAN | NDLING AND RECORDKEEPING | 64 |
| | 9.1. | Case I | Report Forms (CRFs) | 64 |
| | 9.2. | Retent | tion of Records | 64 |
| 10. | QUA | LITY ( | CONTROL AND QUALITY ASSURANCE | 65 |

| 10.1. S | Study Monitoring | 65 |
|---|---|---|
| 10.2. A | Audits and Inspections | 65 |
| 11. ETHIC | S | .66 |
| 11.1. E | Ethics Review | 66 |
| 11.2. E | Ethical Conduct of the Study | 66 |
| 11.3. V | Written Informed Consent | 66 |
| 11.4. Г | Disclosure of Data | 67 |
| 12. REFER | RENCES | 68 |
| | List of Tables | |
| Table 1. I | OHE PK Parameters, mean (±SD); STS101-001, Part 1 | 27 |
| Table 2. I | OHE PK Parameters, mean (±SD); STS101-001, Part 2 | 27 |
| Table 3. L | Laboratory Tests | 36 |
| Table 4. A | Adverse Event Relationship to Study Drug | 54 |
| Table 5. A | Assessment of Adverse Event Severity | 54 |
| | List of Figures | |
| Figure 1. S | STS101 Device | 25 |
| | Dihydroergotamine mesylate chemical structure | |
| _ | Study Schematic | |
| | List of Appendices | |
| Appendix A | A. Schedule of Assessments | 71 |
| Appendix E | 3. List of Allowed and Disallowed Other Headache Types | 72 |
| Appendix C | | |
| Appendix I | D. STS101 Instructions for Use | 75 |
| Appendix E | E. 24-Hour Migraine Quality of Life Questionnaire | 76 |
| Appendix F | F. Headache Impact Test (HIT-6 <sup>TM</sup> ) | 78 |
| Appendix C | G. Sheehan Suicidality Tracking Scale (S-STS) | <del>7</del> 9 |

#### List of Abbreviations and Definitions of Terms

Abbreviation or specialist term Explanation

24-MQoL 24-hour Migraine Quality of Life Questionnaire

AE Adverse Event

ALT Alanine Aminotransferase

ANOVA Analysis of variance

AST Aspartate Aminotransferase

AUC Area Under the Concentration-Time Curve

BMI Body Mass Index
BUN Blood Urea Nitrogen
CBC Complete Blood Count

CGRP Calcitonin Gene-Related Peptide

CM Concomitant Medication

C<sub>max</sub> Maximum Observed Plasma Concentration

CRF Case Report Form

CRO Contract Research Organization

DHE Dihydroergotamine
EC Ethics Committee
ECG Electrocardiogram

eCRF Electronic Case Report Form

e-diary Electronic diary in handheld device
FDA Food and Drug Administration
FIS Functional Impairment Scale

GCP Good Clinical Practice

hCG Human Chorionic Gonadotropin HPMC Hydroxypropyl Methylcellulose

ICF Informed Consent Form

ICHD3 International Classification of Headache Disorder, 3rd Edition

IM Intramuscular IN Intranasal

IRB Institutional Review Board

ITT intent-to-treat
IV Intravenous
max maximum

MBS bothersome symptom
MCC Microcrystalline Cellulose

Abbreviation or specialist term Explanation

MedDRA Medical Dictionary for Regulatory Activities

min minimum

mITT modified intent-to-treat

NOAEL No Observed Adverse Effect Level

PK Pharmacokinetic
PP per protocol

PT Preferred Term (in MedDRA dictionary)

SAE Serious Adverse Event
SAP Statistical Analysis Plan

SC Subcutaneous
SD Standard Deviation

SOC System Organ Class (in MedDRA dictionary)

T<sub>1/2</sub> Terminal Elimination Half-Life

TEAE Treatment Emergent Adverse Events

#### STUDY PROTOCOL REVISION HISTORY

## Changes in Version 1 (May 17, 2021)

Investigational product dose strength: The sponsor decided to conduct this Phase 3 study with the 5.2 mg STS101 dose strength (equivalent to 6.0 mg of DHE mesylate USP) instead of the 8.6 mg dose strength. In all protocol sections all references to the 8.6 mg dose strength have been replaced with the 5.2 mg dose strength.

The sponsor decided to increase the number of study sites to 130. In all protocol sections all references to the number of sites has been updated to 130

#### Synopsis (page 9) and Section 4.2 Subject Exclusion Criteria (page 42)

Added Exclusion Criteria #20:

Score of ≥0 on any of the questions 1-14 of the Sheehan Suicidality Tracking Scale

#### **Rationale:**

FDA requirement to explore treatment emergent suicidal ideation and behavior for drugs in neurological indications.

#### Section 1.2.1 STS101 Device (page 25)

New image of STS101 device without cap was added since the device used in this study will not have a cap.

#### Section 1.3 Summary of Nonclinical Data (page 28)

Minor changes in the text to address higher margins of safety for 5.2 dose strength.

#### Section 1.5 Rationale for Study (page 29)

Minor changes in the text to delete references to 8.6 mg dose strength.

Section 3.2.10 Clinical Laboratory Tests (Table 3, page 36); Section 3.3.3 Randomization Visit (page 38); Section 7.1.2.5 Serum & Urine Pregnancy Test (page 52); Appendix A Schedule of Assessments (page 71)

Added urine pregnancy test conducted at Visit 2.

## Section 3.2.10.1 (page 36) & 7.1.2.7 (page 52) Lab testing for chest related symptoms or adverse events

Added sections to describe additional lab tests for subjects who report chest related symptoms or adverse events.

#### Section 3.2.11 Electrocardiogram (page 36)

Added sections to describe additional ECGs for subjects who report chest related symptoms or adverse events.

Section 3.2.15 Sheehan Suicidality Tracking Scale (page 37); Section 3.3.2 Screening Visit & Period (page 38); Section 3.3.3 Randomization Visit (page 38); Section 3.3.4 Final Visit/Early termination (Visit 3), (page 39); Section 7.1.2.8 Safety Evaluation (page 53); Section 8.3.8.8 Safety Analysis - Sheehan Suicidality Tracking Scale (page 63); Appendix A Schedule of Assessments (page 71); Appendix G Sheehan Suicidality Tracking Scale (page 79)

Added completion of Sheehan Suicidality Tracking Scale at Visits 1, 2 and 3 and analysis of data in safety analysis.

## **Section 4.2 Subject Exclusion Criteria (page 41)**

Added missing words "medication overuse headache" to Exclusion criteria #3

## Section 5.6 Investigative Product Handling & Disposal (page 46)

Minor text edits.

#### Section 8.3.6 Analysis Methods for Efficacy Endpoints (page 61)

Minor text changes.

## Appendix A Schedule of Assessments (page 71)

Minor text change reg. follow up visit window

#### **Appendix D STS101 Instructions for Use (page 75)**

New instructions for use illustration added.

## 1. BACKGROUND INFORMATION

#### 1.1. Introduction

Satsuma Pharmaceuticals, Inc. (Satsuma) is developing STS101 (dihydroergotamine nasal powder), a drug-device combination of a dihydroergotamine (DHE) mesylate dry powder formulation prefilled in a single use delivery device for nasal administration. DHE mesylate is currently indicated for the acute treatment of migraine headaches with or without aura and the acute treatment of cluster headache episodes. DHE mesylate is available as a solution for subcutaneous (SC), intramuscular (IM), or intravenous (IV) administration and as a nasal spray (IN) (D.H.E. 45® Prescribing Information 2017; Migranal® Prescribing Information 2017).

DHE mesylate is a semi-synthetic derivative of ergotamine tartrate that has been used effectively to treat migraine since 1945 (Silberstein 2003) and was first approved in U.S. in 1946. The antimigraine activity of DHE mesylate is likely related to the agonist activity at 5-HT<sub>1B</sub>, 5-HT<sub>1D</sub>, and 5-HT<sub>1F</sub> receptors (Dahlöf 2012). Additionally, DHE mesylate can cause vasoconstriction via CGRP release by stimulating adrenergic  $\alpha_{2A/2c}$  and 5-HT<sub>2A</sub> receptors and may inhibit neurogenic inflammation in peripheral meningeal tissues and nociceptive neuronal transmission centrally in the trigeminal nucleus caudalis (Hoskin 1996; Burstein 2004; Silberstein 2003; Dahlöf 2012; González-Hernández 2018). The DHE mesylate-related side effects of nausea and vomiting are likely related to activation of central 5-HT<sub>1A</sub> receptors and dopamine D<sub>2</sub> receptors (Silberstein 2003).

DHE mesylate is listed as first-line treatment in migraine treatment guidelines from the American Academy of Neurology (Marmura 2015). The effectiveness of DHE mesylate via intravenous, intramuscular, subcutaneous, intranasal and orally inhaled administration routes has been demonstrated (Raskin 1986; Winner 1996; Gallagher 1996; Carleton 1998; Edwards 2001; Aurora 2011). In these studies, treatment with DHE mesylate has consistently resulted in headache relief in 50 to 70% of the treated patients at 2 hours after administration.

However, patient acceptance of DHE mesylate has been limited due to these shortcomings:

- D.H.E.45<sup>®</sup> (Injectable DHE mesylate solution)
  - o Inconvenience and side effects of administration by injection (IV, IM, SC)
  - DHE mesylate-related side effects, especially nausea, which is likely related to rate of administration (IV) and C<sub>max</sub> and has been reported to occur less frequently when plasma concentrations remain below 6-10 ng/mL (Cook 2009)
- Migranal® (DHE mesylate intranasal spray)
  - o Inconvenient multi-step procedure of vial opening, spray device-to-vial assembly, and priming (Migranal® Administration Instructions 2017)
  - o Inconvenient administration procedure requiring four 0.125 mL sprays (two in each nostril, repeated after 15 minutes) (Migranal® Prescribing Information 2017) and Migranal® Administration Instructions 2017)

- Low and variable bioavailability (Tfelt-Hansen 2013; Migranal<sup>®</sup> Prescribing Information 2017)
- o Slow onset of action (Tfelt-Hansen 2013)
- o Drug run off into the pharynx and out of the nose (Djupesland 2013)
- Side effect of bad or altered sense of taste (Migranal<sup>®</sup> Prescribing Information 2017; van der Kuy 1999).

STS101 (DHE nasal powder) is designed and being developed to address the shortcomings of the injectable and intranasal DHE mesylate formulations:

- STS101 is designed to be easy and convenient for patients to quickly self-administer during a migraine attack.
- STS101 is rapidly and consistently absorbed with  $T_{max}$ ,  $C_{max}$  and AUC values falling within ranges that have previously been established to be effective for DHE mesylate.
- Consistent with DHE mesylate effectiveness data reported in multiple studies, STS101 treatment is expected to be effective in early and late treatment of migraines, in attacks with and without allodynia, and to result in high 24-hour pain-free and low 24-hour recurrence rates.

## 1.2. STS101 Description

STS101 is a drug-device combination product consisting of a powder formulation of DHE mesylate prefilled in a single use delivery device for intranasal (IN) administration.

#### **1.2.1.** STS101 Device

STS101 will be delivered by a pre-filled single use device, which is a manually operated and air driven device specifically designed for IN drug delivery (Figure 1).

Figure 1. STS101 Device



#### 1.2.2. STS101 Powder Formulation

STS101 is a white to off-white powder formulation containing DHE mesylate, microcrystalline cellulose (MCC), hypromellose (hydroxypropyl methylcellulose, HPMC), and mannitol.

#### 1.2.2.1. DHE Mesylate Information

DHE mesylate is a semi-synthetic derivative of ergotamine tartrate and is known chemically as ergotaman-3′,6′,18-trione,9,10-dihydro-12′-hydroxy-2′-methyl-5′-(phenylmethyl)-,(5′ $\alpha$ )-,monomethanesulfonate. Its molecular weight is 679.80 and its empirical formula is  $C_{34}H_{41}N_5O_8S$ . The chemical structure is shown in Figure 2.

Figure 2. Dihydroergotamine mesylate chemical structure

#### 1.2.3. DHE Mechanism of Action in the Treatment of Migraine

The antimigraine activity of DHE is likely related to the agonist activity at 5-HT<sub>1B</sub>, 5-HT<sub>1D</sub>, and 5-HT<sub>1F</sub> receptors (Dahlöf 2012). Additionally, DHE can cause vasoconstriction via CGRP release by stimulating adrenergic α<sub>2A/2c</sub> and 5-HT<sub>2A</sub> receptors and may inhibit neurogenic inflammation in peripheral meningeal tissues and nociceptive neuronal transmission centrally in the trigeminal nucleus caudalis (Hoskin 1996; Burstein 2004; Silberstein 2003; Dahlöf 2012; González-Hernández 2018). The DHE mesylate-related side effects of nausea and vomiting are likely related to activation of central 5-HT<sub>1A</sub> receptors and dopamine D<sub>2</sub> receptors (Silberstein 2003). Because of slow diffusion from the receptor biophase, the effects of DHE mesylate last far longer than can be expected from plasma concentrations (Dahlöf 2012; Tfelt-Hansen 2013).

#### 1.2.4. STS101 DHE Pharmacokinetics

In a 2-part, three period, cross-over Phase 1 study, 15 healthy subjects were dosed with ascending doses of 1.3, 2.6 and 5.2 mg STS101 (equivalent to 1.5, 3.0, and 6.0 mg DHE mesylate USP). STS101 demonstrated dose dependent plasma concentrations. Table 1 shows selected PK parameters of Part 1 of the study.

Table 1. DHE PK Parameters, mean (±SD); STS101-001, Part 1

| Parameter | STS101 (1.3 mg) | STS101 (2.6 mg) | STS101 (5.2 mg) |
|---|---|---|---|
| C <sub>max</sub> (pg/mL) | 645 (418) | 1243 (576) | 1870 (823) |
| $T_{max}(h)$ | 0.7 (0.28) | 0.7 (0.47) | 0.4 (0.12) |
| AUC <sub>0-30min</sub> (h*pg/mL) | 188 (137) | 362 (225) | 606 (295) |
| AUC <sub>0-2hr</sub> (h*pg/mL) | 956 (591) | 1683 (719) | 2549 (1132) |
| AUC <sub>0-inf</sub> (h*pg/mL) | 4172 (1860) | 7022 (2557) | 10150 (3814) |
| T <sub>1/2</sub> (h) | 12.9 (2.1) | 12.6 (1.3) | 12 (1.6) |

Source: STS101-001 Data Tables, February 2019

In Part 2 of the study, 27 healthy subjects were dosed with 5.2 mg STS101 (equivalent to 6.0 mg DHE mesylate USP), 1.0 mg IM DHE mesylate, and 2.0 mg intranasal DHE mesylate spray in a randomized order. Table 2 shows selected PK parameters.

Table 2. DHE PK Parameters, mean (±SD); STS101-001, Part 2

| Parameter | IM DHE Mesylate<br>(1.0 mg) | Migranal<br>(IN DHE Mesylate Spray<br>2.0 mg) | STS101<br>(DHE Nasal Powder 5.2 mg<br>(Equivalent to 6.0 mg<br>DHE Mesylate USP) |
|---|---|---|---|
| C <sub>max</sub> (pg/mL) | 3368 (840) | 961 (727) | 2175 (884) |
| T <sub>max</sub> (h) | 0.37 (0.3) | 1.04 (0.4) | 0.6 (0.4) |
| AUC <sub>0-30min</sub> (h*pg/mL)* | 1357 (389) | 152 (131) | 686 (326) |
| AUC <sub>0-2hr</sub> (h*pg/mL)* | 4791 (908) | 1316 (990) | 2979 (1147) |
| AUC <sub>0-inf</sub> (h*pg/mL) | 13650 (2143) | 6498 (3551) | 12030 (4716) |
| T <sub>1/2</sub> (h) | 11.2 (1.93) | 12.7 (2) | 11.8 (2.2) |

Source: STS101-001 Data Tables, February 2019

Additional information including may be found in the STS101 Investigator's Brochure.

## **1.2.5. DHE Clinical Experience**

Migranal® (DHE mesylate intranasal liquid) and D.H.E. 45® (DHE mesylate injectable solution), approved in the United States in 1998 and 1946, respectively, have been prescribed to a large number of patients with migraine headaches. A detailed summary of human experience with marketed DHE mesylate formulations and other data regarding Migranal and DHE mesylate Injectable solution can be found in the STS101 Investigator's Brochure.

## 1.2.6. DHE Mesylate Pregnancy Category

DHE mesylate may cause fetal harm when administered to a pregnant woman. There are no adequate studies of DHE mesylate in human pregnancy, but developmental toxicity has been demonstrated in experimental animals. DHE mesylate possesses oxytocic properties and, therefore, should not be administered during pregnancy. If this drug is used during pregnancy, or if the patient becomes pregnant while taking this drug, the patient should be apprised of the potential hazard to the fetus. DHE mesylate is designated Pregnancy Category X in the U.S (D.H.E. 45® Prescribing Information 2017; Migranal® Prescribing Information 2017).

## 1.3. Summary of Nonclinical Data

The nonclinical toxicology program for STS101 was designed to supplement the known nonclinical studies in support of the general safe use of DHE mesylate. In a GLP 14-day intranasal toxicology study with a 14-day recovery period conducted in dog, the presumed No Observed Adverse Effect Level (NOAEL) of DHE mesylate dose given to dogs (the most sensitive species) was approximately 49-fold more than the planned highest clinical dose of STS101 on a dose/weight (mg/kg) basis and 5-fold more based on a normalized nasal cavity surface area comparison. The results of the dog 14-day study support the presumption that the STS101 DHE mesylate formulation yields no new or unexpected significant toxicity at the highest feasible concentrations possible. The large safety multiples based on the NOAEL provide reassurance that the proposed human clinical dosing is reasonable and safe. The study is summarized in detail in the STS101 Investigator's Brochure.

## 1.4. Summary of Clinical Data for STS101

In the Phase 1 Study STS101-001 (up to 5.2 mg STS101) no serious adverse events occurred and no adverse event led to study or treatment discontinuation. All treatment emergent adverse events recorded were graded as mild, clinically not significant and resolved by the end of the study. As expected, most of the adverse events were local in the nose and described as mild nasal discomfort and taste disturbances usually described as sour or bitter taste. In the Phase 3 Study STS101-002, up to 5.2 mg STS101 showed a favorable safety and tolerability profile. No drug related serious adverse events or deaths occurred during the study. The most common TEAEs were nasal discomfort, dysgeusia, and rhinorrhea. For more details see the STS101 Investigator's Brochure.

## 1.5. Rationale for the study

In the Phase 3 Study STS101-002, STS101 narrowly missed to achieve statistically significant efficacy for the two co-primary endpoints, freedom from pain and most bothersome symptom at 2 hours after use of study medication (Data on file). The main reasons for this were:

- A high rate of severe migraine attacks during the treatment period. Severe migraine attacks are more difficult to treat and tend to have lower response rates for acute migraine treatments (Aurora 2011; Diener 2004). Consistent with the literature severe attacks less response to the study medication.
- The mean delivered dose of study medication was approximately 30% below the label claim because of a combination of suboptimal administration by the study subjects, thicker walls of the pump of the device making it harder to adequately squeeze and some powder loss within the device (Satsuma; Data on file).
- A high placebo response rate in relation to the reported pain and symptom severity of the treated attacks (Aurora 2011; Diener 2004; Dodick 2019; Goadsby 2019; Kuca 2018; Lipton 2019; Tepper 2011)

Satsuma has corrected the device and administration related drug delivery issues, and with these corrections and an increase in sample size, this study is expected to achieve statistically significant efficacy at 2 hours after use of study medication and to demonstrate the clinical benefits of STS101 in the acute treatment of migraine.

This study follows the FDA Guidance<sup>1</sup> and the Guidelines of the International Headache Society for acute migraine studies (Diener 2019) and is being conducted as part of the clinical development program for STS101 to demonstrate the efficacy, safety and tolerability of STS101 in the treatment of acute migraine attacks with or without aura.

<sup>&</sup>lt;sup>1</sup> FDA Guidance for Industry, Migraine: Developing Drugs for Acute Treatment. February 2018.

#### 2. STUDY OBJECTIVES AND PURPOSE

The objectives of this study are:

#### **Primary**

- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from most bothersome symptom at 2 hours after dosing

## Secondary

- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid the use of rescue medication within 24 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve normal function at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 24 hour sustained pain free status
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 48 hour sustained pain free status
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 24 hour sustained freedom from most bothersome symptom status
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve 2 to 48 hour sustained freedom from most bothersome symptom status
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid the use of rescue medication within 48 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid headache pain relapse within 24 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to avoid headache pain relapse within 48 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from most bothersome symptom at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at various timepoints after dosing
- To estimate the probability of a subject to achieve freedom from pain during the 24-hour post dose period
- To estimate the probability of a subject to achieve freedom from the most bothersome symptom during the 24-hour post dose period
- To estimate the probability of a subject to achieve pain relief during the 24-hour post dose period
- To estimate the probability of a subject requiring rescue medication during the 24-hour post dose period

- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from photophobia at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from phonophobia at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from nausea at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from photophobia at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from phonophobia at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from nausea at various timepoints after dosing
- To evaluate the study subject's global impression of the study treatment
- To assess the safety and tolerability of a single dose of 5.2 mg STS101 in the treatment of acute migraine attacks

#### **Exploratory**

- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain and most bothersome symptom by allodynia status at time of dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain and most bothersome symptom at 2 hours after dosing in subjects who wake up with acute migraine attacks
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from pain and most bothersome symptom at 2 hours after dosing in subjects with acute menstrual related migraine attacks
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing in subjects with acute migraine attacks by allodynia status at time of treatment
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing in subjects who wake up with acute migraine attacks
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve pain relief at 2 hours after dosing in subjects with acute menstrual related migraine attacks
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve both, freedom from pain and most bothersome symptom at 2 hours after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve both, freedom from pain <u>and</u> most bothersome symptom at various timepoints after dosing
- To evaluate the efficacy of a single dose of 5.2 mg STS101 to achieve freedom from headache pain and most bothersome symptom (MBS) at 2 hours after dosing by baseline (Visit 2) HIT-6 score
- To evaluate the effects of a single dose of 5.2 mg STS101 on the 24-hour Migraine Quality of Life Questionnaire (24-MQoLQ)

#### 3. STUDY DESIGN

## 3.1. Overall Study Design and Plan

This is a multi-center, single-dose, randomized, double-blind, placebo-controlled, parallel group study in approximately 1400 subjects with acute migraine (ages 18 to 65 years).

After establishing initial eligibility, the study participants will be trained in the use of the electronic diary (e-diary) to record their headache attacks for 15 days during the screening period. Attack pain severity, presence of symptoms (nausea; photophobia, phonophobia) and impact on functional status will be documented.

The study subjects will also be trained in the administration of study medication and use of the STS101 device, and undergo Placebo Response Reduction training, designed to improve discrimination between placebo and drug effects in clinical trials.

After establishing full eligibility, the study participants will be trained in the use of the STS101 device and randomized (1:1) to receive:

- 5.2 mg STS101 (equivalent to 6.0 mg of DHE mesylate USP), or
- Placebo (matching nasal powder)

The randomization will be stratified by the use of migraine prevention medication. After the randomization, the study participants will treat a qualifying migraine attack of at least moderate pain severity with the allocated blinded study medication within 4 hours of the onset of the attack.

The study participants will document the following symptoms of their treated migraine before and over 48 hours after study drug administration in an e-diary: migraine headache pain severity, presence of symptoms (photophobia, phonophobia, nausea), presence of allodynia and functionality status. Headache pain severity and symptom data will be documented immediately before drug administration (time 0), at 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after study drug administration. The subjects must select a most bothersome symptom among photophobia, phonophobia, and nausea immediately before study drug administration.

If subjects require rescue medication, they will be encouraged to wait until the 2-hour post study drug administration data collection timepoint. The use of triptans, other ergot-containing products (including DHE mesylate and ergotamine), lasmiditan, ubrogepant and rimegepant as rescue medications should be avoided for 24 hours after study drug administration. The study participants will return to the study site within approximately one week of the treated migraine attack.

Adverse events, objective nasal evaluation data, safety laboratory data, vital sign data and ECGs will be recorded before and after treatment to evaluate the tolerability and safety of STS101.

Sufficient numbers of subjects will be screened to randomize approximately 1400 subjects in the study. The dropout rate is estimated to be less than 35%. Subjects who withdraw or are withdrawn from the study after dosing will not be replaced. However, in the event that the number of drop-

outs or number of subjects with missing data exceeds initial expectations, subjects who withdraw or are withdrawn might be replaced.

Figure 3 displays the study schematic design:



## 3.2. Study Procedures Descriptions

The following list is a description of the procedures to be completed at screening and during the study:

#### 3.2.1. Informed Consent

An Ethics Committee (EC)/Investigational Review Board (IRB)-approved informed consent form (ICF) must be signed and dated by each study subject prior to any study procedures being performed and a copy must be given to the subject.

## 3.2.2. Assignment of Subject Identification Number

Each subject will be assigned an individual subject identification number. The first three digits will identify the study site (ranging from 001 to 999) and last three digits will identify the subject as a running number starting with 001. As an example, the first subject entering screening at site 001 would receive the subject identification number 001-001, the second subject 001-002 etc.

#### 3.2.3. Inclusion and Exclusion Criteria Assessment

All subjects must qualify for the study based on the inclusion and exclusion criteria specified in Section 4.1 and Section 4.2, respectively.

## 3.2.4. Medical History, Demographics, Concomitant and Prior Medications

A complete medical history will be obtained including a review of all major organ systems, and a history of alcohol, tobacco and caffeine use. Demographics will include gender, date of birth

race, ethnicity, relationship status, employment status and education level. Prior medications will include all medications taken for 28 days prior to Screening. The medical history, demographics and a list of concomitant and prior medications, concomitant procedures and non-drug therapies will be documented at the screening visit (Visit 1).

In female subjects who menstruate the following additional information will be documented for the three months prior to the Screening Visit:

- Timing and duration of menstruation in each month
- Occurrence of migraine headaches on day 1 ( $\pm$  2 days) of menstruation in each month

Previous or current triptan use will be documented. Subjects who have previously or are currently using triptans will be asked to estimate how often they experience(d) pain relief (moderate or severe pain becoming mild to no pain) with triptan use:

• >75% of the time; >50 to 75% of the time; >25 to 50% of the time;  $\le 25\%$  of the time

Medical Records and source documentation to support important diagnoses, e.g., migraine history and inclusion/exclusion criteria must be provided or obtained whenever possible.

## 3.2.5. Headache Impact Test (HIT-6<sup>TM</sup>)

At the Randomization Visit (Visit 2), subjects will complete the 6-question Headache Impact Test (Appendix F), a tool for assessing the impact of headache on daily life in subjects with migraine (Yang 2010).

## 3.2.6. Physical Examination

A physical examination will be performed at Screening (Visit 1), Randomization (Visit 2) and at the Follow-up/early termination visit. The examination will include all major body systems with the exception of genitourinary. Site Personnel performing the physical exams must be qualified by training and licensure.

## 3.2.7. Vital Signs

Vital signs will be obtained at Screening (Visit 1), Randomization (Visit 2), and at the Follow-up/early termination visit. Vital signs will include temperature, sitting blood pressure (to be taken after 5 minutes of sitting), and pulse rate.

## 3.2.8. Weight, Height and Body Mass Index (BMI)

Subjects will be weighed in street clothes after removing shoes, coat or jacket. Weight will be measured at Screening, Randomization, and at the follow-up/early termination visit. Subject height will only be measured at screening, without shoes. Subjects will have their BMI calculated at the Screening visit (Visit 1) using the following formula: BMI = weight (kg)/height (m<sup>2</sup>).

#### 3.2.9. Evaluations of Effects in the Nose

#### 3.2.9.1. Objective Assessment of Nasal Symptoms

This is a 5-item assessment to be completed by a qualified physician, Nurse Practitioner, or physician assistant. Using categorical scales ranging from "none" to "severe", the physician will rate various aspects of the findings on physical examination of the nasal cavity. The questionnaire and detailed instructions for completion are shown in Appendix C.

The Objective Assessment of Nasal Symptoms will be performed during Screening (Visit 1), Randomization (Visit 2), and at the Follow-up/early termination Visit (Visit 3). Assessment sheets must be retained for all subjects. The person performing the assessments should be the same at all visits whenever possible.

## 3.2.10. Clinical Laboratory Tests

A designated central laboratory will perform the hematology, biochemistry, urinalysis and diagnostic tests as specified in Table 3.

Samples for clinical laboratory tests will be taken at Screening (Visit 1) and at the Follow-up/early termination visit (Visit 3). All samples will be collected in accordance with the Study Laboratory Manual and shipped to the designed central laboratory.

Laboratory reports will be reviewed by the investigator and out of range values will be identified and may be repeated at the Investigator's discretion. The Investigator will determine if any out of range values are clinically-significant and require recording as adverse events (AEs) in the electronic Case Report Form (eCRF). All clinically-significant out of range laboratory values obtained at the Randomization Visit or Follow-up visit will be followed until they return to normal or become medically stable.

Laboratory tests with exclusionary results at Visit 1, may be repeated with prior approval by the Medical Monitor. The repeat test should be done at an unscheduled visit (UV) before the subject returns for the randomization visit (Visit 2).

**Table 3.** Laboratory Tests

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| Hematocrit Hemoglobin MCV Red Blood Cell Count Platelet Count White Blood Cell Count (with Differential) | Albumin Alkaline Phosphatase Alanine Transaminase (ALT) Aspartate Transaminase (AST) Blood Urea Nitrogen (BUN) Calcium Chloride Cholesterol profile Creatine phosphokinase Creatinine Gamma Glutamyl Transferase Glucose Lactate Dehydrogenase Potassium Sodium Direct and Total Bilirubin Total Protein Thyroid function tests (TSH, total T3 & T4) FSH Serum pregnancy test | Appearance Color pH Specific Gravity Protein Glucose Ketones Occult Blood Nitrites Urobilinogen Leukocytes Bilirubin Urine microscopy, if necessary |
| | Diagnostic Screening | |

#### Urine

Alcohol & Drug Panel, including Amphetamines, Cannabinoids, Cocaine, Opiates, PCP and Methadone

#### **Urine Pregnancy test**

To be performed at Visit 2 on all females regardless of childbearing potential Test kits will be provided by central laboratory.

#### 3.2.10.1. Lab Testing for Chest Related Symptoms or Adverse Events

In subjects who report chest related symptoms or adverse events, the following markers should be evaluated (if symptoms are reported to the site within 48 hours of onset): total creatine kinase (CK), CK-myocardial band (CK- MB), aspartate aminotransferase (AST), lactate dehydrogenase (LDH), cardiac troponins (Troponin T; Troponin I), and myoglobin. A blood sample for analysis of DHE plasma concentration should also be drawn.

## 3.2.11. Electrocardiogram

A 12-lead ECG will be performed at Screening (Visit 1) and at the Follow-up/early termination Visit (Visit 3). The investigator or a qualified delegate will review the ECG to assure subject eligibility. All ECGs will be done in triplicate approximately one minute apart.

In subjects who report chest related symptoms or adverse events, an ECG (in triplicate) should be recorded if symptoms are reported to the site within 48 hours of onset.
### 3.2.12. Adverse Events Recording

Adverse events will be recorded and assessed as specified in Section 7.

### 3.2.13. Electronic Headache Diary

Study participants will receive a handheld device for collection of data in an electronic diary. At the Screening and Randomization Visits, study participants will receive training in the use of the device and completion of the diaries. During the screening period the study participants will document their headaches for 15 days. Headaches and migraine attacks (including information on pain severity and symptoms) will be documented.

During the treatment period, the study participants will document sign and symptoms identifying a migraine headache, the pain severity of their treated migraine attack, presence and severity of symptoms (photophobia, phonophobia, nausea, allodynia) and functional status over the 48-hour period after study drug administration in the e-diary.

The complete content and the training procedures for the electronic diary device will be described in separate documents.

### 3.2.14. Placebo Response Reduction Training

At Visit 1 and Visit 2, study participants will undergo a Placebo Response Reduction (PRR) Training that consists of a set of subject and staff educational materials for training on appropriate expectations of personal benefit while participating in a clinical trial and to neutralize excessive expectations that drive high placebo responses in clinical trials.

The complete content and the PRR training procedures will be described in separate documents.

### 3.2.15. Sheehan Suicidality Tracking Scale (S-STS)

All study subjects will complete the Sheehan Suicidality Tracking Scale (S-STS) (Appendix G) at Visits 1, 2 and 3.

### 3.3. Schedule of Observations and Procedures

Appendix A shows the procedures for the study. The following assessments should be completed at the designated time period(s).

### 3.3.1. Screening Procedures

Initial screening will be performed at Study Entry, and it will determine whether subjects will qualify for the study.

### 3.3.2. Screening Visit & Period (Day-30 to Day -1)

Subject screening procedures and study entry procedures include:

- a. Signing of informed consent
- b. Review of inclusion/exclusion criteria
- c. Recording of demographic data
- d. Medical history, including migraine history, concomitant medications, procedures and non-drug therapies
- e. Physical examination
- f. Vital signs (including pulse rate, sitting blood pressure and temperature)
- g. Body weight, height and BMI calculation
- h. Objective Assessment of Nasal Symptoms
- i. Completion of Sheehan Suicidality Tracking Scale
- j. STS101 device training
- k. Electronic device & diary use training
- 1. Placebo response reduction training
- m. Clinical laboratory tests
- n. Urinalysis
- o. Serum pregnancy test (all female subjects)
- p. Urine drug and alcohol screen
- q. 12-lead ECG (in triplicate)
- r. Adverse event recording
- s. Completion of Headache Diary by subject (for 15 days within screening period)

### 3.3.3. Randomization Visit (Visit 2; Day1)

- a. Review of Headache diary data
- b. Vital signs (including pulse rate, sitting blood pressure and temperature)
- c. Physical examination
- d. Weight
- e. Review of concomitant medications, procedures and non-drug therapies
- f. Serum pregnancy test (all female subjects)
- g. Urine pregnancy test (all female subjects)
- h. Objective Assessment of Nasal Symptoms
- i. Completion of Sheehan Suicidality Tracking Scale
- j. Completion of HIT-6 instrument

### k. Review of eligibility criteria

Any subject that no longer qualifies for study participation based on findings in any of the procedures will be withdrawn from the study as a screen failure and the reasons recorded on the screen failure log.

If the subject still meets all eligibility criteria for study participation, the following procedures will be done:

- a. Randomization
- b. STS101 device and administration training
- c. Dispense Investigational Product
- d. Electronic device and diary use training
- e. Placebo response reduction training

The subject has 56 days to treat a qualifying migraine attack in the Treatment Period.

### 3.3.4. Final Visit/Early Termination (Visit 3)

Subjects will undergo final safety assessment procedures within approximately one week (7 days  $\pm$  3 days) after use of study medication. If a subject has not treated a qualifying migraine within 56 days of randomization, the subject should return to the site and all final visit procedures should be performed.

The follow-up visit/early termination procedures will comprise the following:

- a. Physical examination
- b. Vital signs (including pulse rate, sitting blood pressure and temperature)
- c. Review of concomitant medications, procedures and non-drug therapies
- d. Serum pregnancy test (all female subjects)
- e. Clinical laboratory tests
- f. Urinalysis
- g. 12-lead ECG (in triplicate)
- h. Completion of Sheehan Suicidality Tracking Scale
- i. Objective Assessment of Nasal Symptoms
- j. Patient Subjective Impression Questions (see Section 6.2)
- k. Adverse event recording
- 1. Collect used Investigational Product (STS101 device)
- m. Collect electronic diary device

### 4. SELECTION AND WITHDRAWAL OF SUBJECTS

A total of approximately 1400 adult male and female subjects aged 18 to 65 years with acute migraine headaches will be randomized.

### 4.1. Subject Inclusion Criteria

A subject will be eligible for inclusion in this study only if all of the following criteria applied:

- 1. English speaking males or females, 18-65 years of age at the time of Screening Visit
- 2. Signed Informed Consent Form
- 3. Subject has at least 1-year history of migraines (with or without aura), according to the International Classification of Headache Disorder, 3rd Edition (ICHD3), including the following:
  - a. Migraine onset before the age of 50 years
  - b. Migraine attacks, on average, lasting 4-72 hours if untreated
  - c. Migraine headache frequency of 2 to 8 attacks of moderate or severe pain intensity per month in each of the 3 months prior to the Screening Visit
  - d. Fewer than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit
  - e. Individual migraine attacks separated by at least 2 days of no headache pain
  - f. Subject is able to distinguish migraines from other headache types, e.g., tension-type or cluster headache.
- 4. Subjects on preventive migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to study entry and have no plans to change the dose during the study
- 5. Female subjects will be included if they are post-menopausal (at least 1 year since last menses) or surgically sterilized; or if they are of childbearing potential, they are not breastfeeding, have a negative pregnancy test, have no intention of becoming pregnant during the course of the study, and are using adequate contraceptive drugs or devices during the course of this study. Medically acceptable methods of contraception that may be used by the subject and/or her partner are:
  - a. Simultaneous use of male condom and intra-uterine contraceptive device placed at least 4 weeks prior to screening (Visit 1)
  - b. Simultaneous use of male condom with intravaginally applied spermicide and diaphragm
  - c. Simultaneous use of male condom and hormonal contraceptives started at least 4 weeks prior to screening (Visit 1)
  - d. Surgical sterilization of their partner(s) at least 6 months prior to screening (Visit 1)

- 6. Intact nasal mucosa (Appendix C, Objective Assessment of Nasal Symptoms: no ulceration; no bleeding; no or mild erythema; no or mild swelling; and no or mild rhinorrhea), and no other nasal conditions that may interfere with intranasal dosing at randomization (Visit 2)
- 7. Willing and able to comply with the requirements of the protocol and follow directions from the clinic staff
- 8. Adequate compliance (≥80%) in the completion of the e-diary during the Screening Period

# 4.2. Subject Exclusion Criteria

- 1. Pregnant or breast-feeding women
- 2. Women of child-bearing potential not using or not willing to use highly effective contraception
- 3. Diagnosis of headache conditions other than migraine with or without aura, including diagnosis of basilar or hemiplegic migraines, medication overuse headache or cluster headache
- 4. Abnormal physical findings of clinical significance which would interfere with the objectives of the study at the screening or randomization visit examination
- 5. History of coronary artery disease, coronary artery vasospasm (including Printz-metals' angina), clinically significant arrhythmia or, peripheral vascular disease, ischemic disease (e.g., Raynaud's syndrome, ischemic bowel syndrome, angina pectoris, myocardial infarction, or documented silent ischemia); percutaneous coronary intervention, or cardiac surgery
- 6. History of cerebrovascular disease, including but not limited to stroke, transient ischemic attack, cerebral hemorrhage, subarachnoid hemorrhage
- 7. Presence of two or more of the following cardiovascular risk factors:
  - a. Previous diagnosis of hypertension or currently taking antihypertensive medication
  - b. Previous diagnosis of hypercholesteremia, or currently taking cholesterol lowering treatment or LDL >159 mg/dL at screening (Visit 1; note: re-draws prior to Visit 2 may be permitted)
  - c. Obesity (BMI > 31)
  - d. Diabetes mellitus
  - e. Family history of premature coronary artery disease (in male first-degree relatives < 55 years or female first-degree relatives < 65 years)
  - f. Females who are surgically or physiologically postmenopausal
  - g. Males 46 or older
- 8. Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at screening (Visit 1; note: re-draws prior to Visit 2 may be permitted)
- 9. Severely impaired hepatic function (liver function tests ALT or AST greater than 2 times upper limit of normal) or renal function (serum creatinine greater than 1.5 times the upper limit of normal) at screening (Visit 1; note: re-draws prior to Visit 2 may be permitted)

- 10. Screening 12-lead ECG showing any clinically significant abnormalities at screening (Visit 1)
- 11. Systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, at screening (Visit 1)
- 12. Diagnosis of major depression with current symptoms, psychosis, alcohol abuse or dependence, drug abuse or dependence, major psychiatric conditions (e.g., schizophrenia, psychosis or Bipolar disorder), or dementia. Other significant neurological or psychiatric disorders (including other pain syndromes or risk of suicide) that in the opinion of the investigator might interfere with study participation and assessments or subject safety
- 13. Any clinically significant symptoms or conditions, including but not limited to central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator might interfere with study assessments or subject safety
- 14. Participation in another drug research study within 30 days of Screening Visit or within less than 5 half-lives of tested drug (whichever is longer)
- 15. Concomitant use of potent CYP3A4 inhibiting medications, for example protease inhibitors (e.g., ritonavir, nelfinavir, indinavir, saquinavir, tipranavir, lopinavir, atazanavir, darunavir), macrolide antibiotics (e.g., erythromycin, clarithromycin, troleandomycin), or strong imidazole antifungals (e.g., ketoconazole, and itraconazole)
- 16. Previously shown hypersensitivity to ergot alkaloids or the inactive ingredients of STS101 (microcrystalline cellulose, hydroxypropyl methylcellulose, mannitol)
- 17. Concomitant use of more than one preventive migraine medication
- 18. Current use of opioids, or cannabis or cannabinoid containing products
- 19. Concomitant use of peripheral and central vasoconstrictors including but not limited to amphetamines, phenylephrine, pseudoephedrine, propranolol and nicotine (from smoking, vaping or smokeless products)
- 20. Score of >0 on any of the questions 1-14 of the Sheehan Suicidality Tracking Scale

# 4.3. Subject Withdrawal Criteria

Subjects will be informed that they are free to withdraw from the study at any time. The Investigator or the Medical Monitor may exercise his/her medical judgment to terminate a subject's participation in the study due to compliance, medical or other reasons. All data normally collected at completion of the study (Visit 3) must be collected as soon as possible once a subject is withdrawn. The primary reason for discontinuation of treatment should be noted in the CRF and source data using the following categories:

a. **Adverse Event:** The subject has experienced an AE that, in the opinion of the Investigator, requires early termination. If a subject is discontinued from the study due to an AE, the Investigator is required to follow the subject until the AE is resolved, or declared medically stable or the subject is lost to follow up.

- b. **Non-compliance:** The subject did not adhere to protocol requirements in a fashion that would impair the data integrity or subject safety.
- c. Withdrawal of Consent: The subject wishes to withdraw from the study.
- d. **Death.** The event causing the death will be an SAE and will be documented.
- e. **Investigator Discretion:** In the Investigator's judgment, continued participation in the study would not be in the best interest of the subject or the study.
- f. **Study Termination:** The Sponsor, or IRB terminates the study.
- g. Lost to follow up. Every effort should be expended to contact the subject and have them return for follow up assessments and return of Investigational Product (used or unused) and the electronic diary device.
- h. **Other:** If subject is discontinued from the study for any reason not applicable to the reasons stated above, this category should be used. The specific reason should then be indicated in the subject's source documents and the appropriate CRF.

### 5. TREATMENT OF SUBJECTS

# 5.1. Description of Investigational Product and Packaging

STS101 is a drug-device combination product consisting of a powder formulation of DHE mesylate prefilled in a single use delivery device for IN administration. The STS101 drug constituent contains a formulation of DHE mesylate, microcrystalline cellulose, mannitol and HPMC. STS101 Placebo consists of the same inactive ingredients but without DHE mesylate.

DHE mesylate is a white or almost white to faintly red powder or colourless crystals. DHE mesylate is known chemically as ergotaman-3′,6′,18-trione,9,10-dihydro-12′-hydroxy-2′-methyl-5′-(phenylmethyl)-,(5′ $\alpha$ )-,monomethanesulfonate. Its molecular weight is 679.80 and its empirical formula is C<sub>34</sub>H<sub>4</sub>1N<sub>5</sub>O<sub>8</sub>S. Further information can be found in the Investigator's Brochure.

The investigational product will be made available as:

- 5.2 mg STS101 dose strength (equivalent to 6.0 mg DHE mesylate USP) as unit dose in a labeled foil wrap.
- Matching placebo as unit dose in a labeled foil wrap.

The non-investigational product will be made available for training during the Screening and Randomization Visits:

- STS101 Empty Training Devices (empty STS101 Device).
- STS101 Filled Training Devices (STS101 Device containing microcrystalline cellulose).

# 5.2. Investigational Product Labeling

The foil wrap will be labeled with a label designating:

- STS101 dose strength (5.2 mg DHE, or placebo)
- Protocol number
- Lot number
- Kit Number
- Name and address of study sponsor
- Recommended storage conditions
- Investigational use only
- Directions: Use as directed following the Instructions for Use
- Warning: For nasal use only
- Blank spaces for: Date dispensed & Subject Number (to be completed by site personnel at time of dispensing)

# 5.3. Investigational Product Storage

Investigational Product supplies are to be stored under secure conditions in a dry, locked, limited access cabinet, at controlled room temperature. All Investigational Product must be stored at room temperature ( $2^{\circ}-30^{\circ}$  C or  $36^{\circ}-86^{\circ}$ F).

The study site pharmacist or designee will maintain an inventory and acknowledge receipt of all shipments of the Investigational Product. Accurate storage and dispensation records must be kept for drug accountability. Supplies of the investigational products will be checked and accountability records will be reviewed at each monitoring visit. A copy of all completed drug accountability forms will be collected by the monitor.

# 5.4. Investigational Product Administration & Training

STS101 will be self-administered by the subjects using the delivery device according to the Instructions for Use.

At Screening (Visit 1) and Randomization (Visit 2), study personnel will train the subject in the study drug preparation and administration. Instructions for Use (Appendix D), an instructional video, STS101 Empty Training Devices and STS101 Filled Training Devices will be used for training of the study subject at both visits.

When using the study medication at home, the study subject will record the following information in the electronic diary:

- Time of dosing (defined as time of last intranasal delivery device actuation).
- The nostril (right or left) into which study drug was administered.
- Whether or not there was any sneezing and/or nose blowing, within 30 minutes after dosing.

Subjects will be instructed to:

- Place clear Cap, Nozzle's Tab and Nasal Device into the plastic bag provided.
- Place the plastic bag and Foil wrap into the carton.
- Return the carton to the clinical site.

# 5.5. Investigational Product Accountability

The Investigational Product will be prescribed by a licensed medical doctor.

The Investigator must maintain accurate records accounting for the receipt and dispensing of the investigational materials. This should consist of a dispensing record including the identification of the person to whom the drug is dispensed, the quantity and the date of dispensing, and the return of study drug/devices.

All Investigational Products dispensed to and taken by subjects must be accurately recorded on an appropriate drug accountability record maintained at the site and reviewed by the study monitor.

All Investigational Products designated for this clinical study must not be administered to any subjects other than those enrolled in this study and may not be utilized for any laboratory or animal research.

## 5.6. Investigational Product Handling and Disposal

Site study staff will retain used and unused Investigational Product at the study site. All used and unused Investigational Product will be reconciled by the Sponsor's designee. All used and unused STS101 devices will be returned to the Sponsor or a designee or if requested by sponsor, destroyed at the study site in compliance with the rules and regulations set forth by the institution conducting the study, and in observance with the rules and regulations of federal agencies concerning prescription only drug products.

# 5.7. Concomitant Medications & Migraine Treatments

Use of any concomitant medications will be documented and reported.

Triptans, ergot alkaloids, Lasmiditan, ubrogepant and rimegepant are not allowed within 48 hours before and for 24 hours after study drug administration.

No other medication intended for treatment of the acute migraine attack should be taken within 24 hours before and for 2 hours after study drug administration.

The concomitant use of more than one prevention medication for migraine is not allowed.

The use of external neuromodulation devices for treatment of acute migraine (e.g., transcutaneous electrical nerve stimulation, transcranial magnetic stimulation) is **not allowed for 48 hours before and 24 hours after study drug administration.** 

If a subject does not experience relief from migraine headache at 2 hours after study medication administration (and after the 2-hour assessments have been completed in the eDiary), the use of the following rescue medication is allowed: aspirin, acetaminophen, NSAIDs, neuroleptics, corticosteroids, antiemetics, muscle relaxants, sedatives, sleep medications, gabapentin.

The concomitant use of potent CYP3A4 inhibiting medications, for example protease inhibitors (e.g., ritonavir, nelfinavir, indinavir, saquinavir, tipranavir, lopinavir, atazanavir, darunavir), macrolide antibiotics (e.g., erythromycin, clarithromycin, troleandomycin), or strong imidazole antifungals (e.g., ketoconazole, and itraconazole) is not allowed.

The chronic daily concomitant use of a peripheral and central vasoconstrictive medication (e.g., amphetamine, methamphetamine, epinephrine) is not allowed. Subjects may use vasoconstrictive medication on a PRN basis, but the use of vasoconstrictive medication is **not allowed within 48** hours before and for 24 hours after study drug administration.

The concomitant use of opioids, or cannabis or cannabinoid containing products is not allowed.

The use of nasal preparations containing decongestants is not allowed within 12 hours before study drug administration.

Further details of allowed and disallowed concomitant medications will be provided in a separate document.

### **5.8.** Treatment Compliance

All used or unused Investigational Product will be returned to the site at Visit 3 at which time the dispensed Investigational Product will be reconciled in the drug accountability log.

# 5.9. Randomization and Blinding

## 5.9.1. Subject Randomization

After evaluation of the subject eligibility and confirmation that subject meets the Inclusion and Exclusion criteria at the Randomization Visit, a study subject will be randomized in the IWRS system according to the pre-programmed randomization schedule. The randomization will be stratified for the use of migraine prevention medication. The randomization process will be described in a separate document.

# 5.9.2. Blinding

The study is a double-blind study of STS101 and matching placebo. No personnel directly involved with the conduct of the study will have knowledge of a subject's treatment assignment. This includes all personnel at the study site, at the sponsor and any CRO involved in the conduct and monitoring of the study. A randomization code will be generated by a statistician independent of the study and not be available to the analysis team until the clinical and data collection, entry, and cleaning processes are complete and database is locked for unblinded analysis.

# 5.9.3. Unblinding Procedures

Unblinding procedures will be described in a separate document.

### 6. ASSESSMENT OF EFFICACY

# 6.1. Efficacy Evaluation Parameters (e-Diary)

The following efficacy evaluation parameters will be programmed in an electronic handheld device (e-Diary) that the study subjects will use to provide their information.

### **6.1.1.** Migraine Headache Pain Severity

The study participants will be prompted to document the pain severity of the treated migraine attack by this request: "Please rate the pain severity of your current migraine headache."

The subject's rating will be documented on a four-point scale from no pain (=0), mild pain (=1), moderate pain (=2) to severe pain (=3).

Headache pain severity ratings will be collected at the onset of the migraine attack, immediately before drug administration (time 0), at 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after study drug administration.

### **6.1.2.** Most Bothersome Symptom

The study participants will be prompted to document the presence of three symptoms, photophobia, phonophobia and nausea during the treated migraine attack by these requests:

For photophobia: "Do you have sensitivity to light?"
For phonophobia: "Do you have sensitivity to sound?"

For nausea: "Do you have nausea?"

For each of the three symptoms, the subject will respond with "Yes" (if symptom present) or "No" (if symptom absent).

Immediately before study drug administration (time 0), the study subjects will be prompted to declare the most bothersome symptom among the symptoms present by this request: "Please indicate which of the symptoms that you have at (sensitivity to light, sensitivity to sound or nausea) bothers you the most at this time."

The presence of the three symptoms will be recorded at the onset of the migraine attack, immediately before drug administration (time 0), at 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after study drug administration.

# **6.1.3.** Evaluation of Allodynia

The presence of allodynia (painful cutaneous sensations) will be assessed by prompting the study subjects to respond to these questions (Ashkenazi 2007; Tepper 2011):

- 1. Is your scalp tender to touch?
- 2. Does combing your hair bother you?

- 3. Does wearing your glasses or sunglasses bother you?
- 4. Does washing your face bother you?
- 5. Are your teeth and gums tender to touch?
- 6. Is your skin over the face tender to touch?

For each question, the possible responses are "Yes", "No" and for questions 2 and 3 also "Not applicable (NA)".

Study subjects answering "Yes" to at least 2 questions will be considered to have allodynia. The presence of allodynia will be assessed immediately before drug administration (time 0), at 2 and 4 hours after study drug administration.

### **6.1.4.** Use of Rescue Medication

Rescue medication is defined as any medication taken to treat the migraine headache after study drug administration.

Any use of medications to treat the migraine headache will be recorded for 48 hours after study drug administration. Study subjects will be encouraged to avoid use of any rescue medication until the 2-hour post study drug administration data collection timepoint.

#### 6.1.5. Evaluation of Function

### **6.1.5.1.** Functional Impairment Scale

The study subjects will be prompted to record their functional status using the Functional Impairment Scale (FIS): "Please rate how much your current migraine headache impacts your ability to function right now."

The subject's rating will be documented on a four-point scale from no impairment (= 0; able to function normal), mild impairment (= 1; able to perform all activities of daily living but with some difficulty), moderate impairment (= 2; unable to perform certain activities of daily living) to severe impairment (= 3; unable to perform most to all activities of daily living or requiring bed rest).

The FIS will be recorded at the onset of the migraine attack, immediately before drug administration (time 0), at 1, 2, 4, 24, and 48 hours after study drug administration.

# 6.1.5.2. 24-hour Migraine Quality of Life Questionnaire

The study subjects will be prompted to complete the 24-hour Migraine Quality of Life Questionnaire (24-MQoL) (Appendix E) at 24 hours after drug administration.

# 6.2. Patient Subjective Impression Questions (Office; Visit 3)

# **6.2.1.** Patient Global Impression

The study subjects will be asked to rate the global impression of the study treatment at Visit 3 with this question: "What is your global impression of the study treatment?"

The subject's rating will be documented on a five-point verbal Likert scale with these response options: very good, good, no opinion, poor, very poor.

# **6.2.2.** Ease of Use Impression

The study subjects will be asked to rate the ease of use of the study medication at Visit 3 with this question: "How easy was the administration of the study medication?"

The subject's rating will be documented on a five-point verbal Likert scale with these response options: very easy, easy, no opinion, not easy, not easy at all.

### 6.2.3. Patient Likelihood of Use

The study subjects will be asked to rate the likelihood of using the study medication at Visit 3 months with this question: "How likely is it that you would use the study medication to treat your migraine if it were available?"

The subject's rating will be documented on a five-point verbal Likert scale with these response options: very likely, likely, no opinion, unlikely, very unlikely.

# 6.2.4. Comparison of study medication with previously used migraine medication

The study subjects will be asked to compare the effects of the study medication with their previously used migraine medication at Visit 3 with answers to these four statements:

Compared to my previous migraine medication, STS101 (the study medication)

- 1. Allows me to return to normal faster
- 2. More consistently treats my migraine
- 3. Works faster
- 4. Keeps migraine from coming back

The answer options for all four statements are: strongly agree; agree; neutral; disagree; strongly disagree.

### 7. ASSESSMENT OF SAFETY

# 7.1. Safety Parameters

The following evaluations and assessments will be conducted during the course of the study (Refer to the Schedule of Assessments in Appendix A).

### 7.1.1. Examinations

### 7.1.1.1. Physical Examinations

A physical examination will include the following body systems: HEENT, Lymphatic, Cardiovascular, Respiratory, Gastrointestinal, Dermatologic, Musculoskeletal, Neurologic and Other.

New physical examination observations that meet the definition of an AE will be recorded on the AE form.

### 7.1.1.2. Height, Weight, and BMI

Subjects will be weighed in street clothes after removing coat or jacket and shoes at the Screening Visit, Randomization visit, and follow-up or early termination visit. At the Screening Visit, subject height will be measured without shoes. Subjects will have their BMI calculated using the following formula: BMI = weight (kg)/height (m<sup>2</sup>).

### **7.1.1.3.** Vital Signs

Vital signs consist of the subject's resting sitting blood pressure, pulse rate, and temperature.

The subject should rest for at least 5 minutes prior to recording the vital signs. The Investigator will review the vital signs and comment on all clinically-significant abnormalities.

### 7.1.1.4. Objective Nasal Symptom Assessments

An assessment of the objective nasal symptoms (Appendix C) will be performed at the Screening, Randomization and follow-up visits.

### 7.1.1.5. Electrocardiogram (ECG)

Standard 12-lead ECG will be performed in triplicate. All ECGs will be reviewed by a competent physician who will comment on any abnormal findings. Clinically significant findings if found at screening or randomization may be a reason to exclude the subject.

### 7.1.2. Laboratory Assessments

Central laboratory tests results will be reviewed for any clinically significant abnormalities by a qualified physician or physician assistant. If any clinically significant findings are present at screening, the subject will be considered a screen failure and ineligible for study participation.

### 7.1.2.1. Hematology

Complete blood count (CBC) with differential including: white blood cell count with differential, red blood cell count, hemoglobin, hematocrit, MCV, and platelet count.

### 7.1.2.2. Serum Chemistry

Serum chemistry including: albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin (direct and total), blood urea nitrogen (BUN), calcium, chloride, cholesterol profile, creatine phosphokinase, creatinine, gamma glutamyl transferase, glucose, lactate dehydrogenase, potassium, sodium, thyroid function tests (TSH, total T3 & T4), and total protein.

### **7.1.2.3.** Urinalysis

Urinalysis examination including: Appearance, color, pH, specific gravity, protein, glucose, ketones, occult blood, nitrites, urobilinogen, leukocytes, bilirubin and if necessary, urine microscopy.

### 7.1.2.4. Urine Drug Screen

Alcohol & Drug Panel: Amphetamines, Barbiturates Benzodiazepines, Cannabinoids, Cocaine, Opiates, PCP and Methadone.

### 7.1.2.5. Serum & Urine Pregnancy Test

A serum HCG pregnancy test will be performed at screening, randomization and the follow-up/early termination visits in all female subjects regardless of child bearing potential. A urine pregnancy test will be performed on all female subjects, regardless of child bearing potential at randomization (Visit 2).

#### **7.1.2.6. Serum FSH test**

A serum FSH test will be performed for any woman who is either surgically menopausal (absence of both ovaries) or physiologically menopausal.

### 7.1.2.7. Lab testing for chest related symptoms or adverse events

In subjects who report chest related symptoms or adverse events, the following markers should be evaluated (if symptoms are reported to the site within 48 hours of onset): total creatine kinase

(CK), CK-myocardial band (CK-MB), aspartate aminotransferase (AST), lactate dehydrogenase (LDH), cardiac troponins (Troponin T; Troponin I), and myoglobin. A blood sample for analysis of DHE plasma concentration should also be drawn.

### 7.1.2.8. Sheehan Suicidality Tracking Scale

The S-STS is a 16-item scale that assesses the seriousness of suicidality risk using a 5-point Likert scale from "not at all" (0) to "extremely" (4) (Sheehan, 2014). The S-STS wil be completed by all subjects at Visits 1, 2 and 3.

### 7.2. Adverse Events

An adverse event (AE) is defined as: "Any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment." An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not related to the investigational product. Treatment emergent adverse events (TEAE) are defined as adverse events recorded after dosing of the investigational product.

AEs will be recorded as volunteered by the subject or solicited through indirect questioning.

AE collection will begin following the subject's signing the informed consent at the Screening Visit (Visit 1) and continue until the follow-up/early termination visit. AEs related to the administration of inactive powder during the administration training at Visit 1 and Visit 2 will also be recorded.

AEs will be solicited at the times indicated in the schedule of assessments by asking a question such as: "Since you were last seen, have you felt unwell or different from usual in any way?" AEs may also be reported spontaneously.

Each AE should be recorded to represent a single diagnosis. Accompanying signs (including abnormal laboratory values) or symptoms related to a single diagnosis should NOT be recorded as additional AEs. If a diagnosis is unknown, sign(s) or symptom(s) should be recorded as an AE(s). Changes in laboratory values are only considered to be AEs if they are judged to be clinically significant (i.e., if some action or intervention is required or if the Investigator judges the change to be beyond the range of normal physiological fluctuation). If abnormal laboratory values are the result of pathology for which there is an overall diagnosis (e.g., increased liver enzymes in hepatitis), the diagnosis only should be reported as an AE.

Any adverse events, signs, and symptoms will be fully recorded on the AE form including date of onset, date of resolution, frequency, severity, seriousness, relationship to the drug, treatments administered and outcome. AEs may also be reported spontaneously at any time.

All AEs must be recorded in the source data and the CRF. Any ongoing AE will be followed, whenever possible, until it resolves, or returns to the baseline condition, or is declared medically stable with no further change expected or the subject is lost to follow up.

# 7.2.1. AE Relationship to Study Drug

An AE will be considered 'related" or "not related" to the use of the investigational product based on the criteria listed in Table 4. Assessment of the causal relationship between any Serious Adverse Event (SAE) and study drug administration will be performed by both the Investigator and the Sponsor. If at least one of the parties assesses the event as related, it will be reported expeditiously as required to the appropriate authorities.

Table 4. Adverse Event Relationship to Study Drug

| Related: | There is "a reasonable possibility" that the event may have been caused by the product under investigation (i.e., there are facts, evidence, or arguments to suggest possible causality). Individual AE reports will be considered "related" to the use of the product if the "not related" criteria are not met. |
|---|---|
| | ernena are not met. |
| Not<br>Related: | There is an unlikely temporal relationship between administration of the product and the onset of the AE (i.e., the event occurred either before, or too long after administration of the product for it to be considered product-related); |
| | The causal relationship between the product, and the AE is biologically implausible (i.e., injury in an automobile accident); |
| | There is a clearly more likely alternative explanation for the AE (i.e., typical adverse reaction to a concomitant drug and/or typical disease-related event). |

# 7.2.2. Assessment of Adverse Event Severity

Table 5 shows the guidelines for rating severity of AEs may be used:

**Table 5.** Assessment of Adverse Event Severity

| Mild: | Awareness of signs or symptoms, but easily tolerated; are of minor irritant type; no loss of time from normal activities; symptoms would not require medication or a medical evaluation; signs and symptoms may be transient, disappearing during continued treatment with study medication. |
|---|---|
| Moderate: | Discomfort enough to cause interference with or modification of usual activities. |
| Severe: | Incapacitating, with inability or notable impairment in work or usual activities; signs and symptoms may be of systemic nature or require medical evaluation; the study drug may be stopped, and treatment for the event may be required. |

### 7.2.3. Serious Adverse Events (SAEs) Recording and Reporting

The Investigator must decide whether each AE meets the definition of an SAE. An SAE is any untoward medical occurrence that at any dose:

- 1. Results in death.
- 2. Is life-threatening.
- 3. Requires inpatient hospitalization or prolongation of existing hospitalization.
- 4. Results in persistent or significant disability/incapacity.
- 5. Is a congenital anomaly/birth defect.
- 6. Is considered medically significant by the Investigator or requires intervention to prevent any one of the outcomes above.

For fatal events, the cause of death is reported whenever known. If an autopsy was performed, an autopsy report should be provided. Death should be reported as the outcome of a specific SAE.

Life-threatening, in the definition of serious, refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.

Reports for hospitalization of elective procedures do not need to be reported as SAEs if there are no precipitating signs/symptoms or worsening of the pre-existing condition that necessitated the procedure. However, SAEs must be reported for any medical complications that prolonged the hospitalization.

Medically significant events are those events considered important in the Investigator's opinion that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above. These will also usually be considered serious.

Any SAE will be reported within 24 hours of knowledge by the Investigator. Investigator should not delay reporting while waiting for clarification or supporting medical information.

The Investigator must complete the required information fields for SAE documentation and reporting in the electronic CRF (AE eCRF and SAE eCRF) and provide any supportive documents available (hospital summaries, diagnostic test results, laboratory test results, etc.). Any subject identifying information must be redacted prior to uploading. The investigator should not wait for these supporting documents in order to notify the medical monitor if doing so would place the notification outside the 24-hour window. All SAEs will also be reported on the AE eCRF and SAE eCRF and concomitant medications (CM) administered in association with the serious AE will be documented on the CM eCRF.

For any information not available at the time of the first report that becomes available later, the Investigator should add this information to both the source documentation and the initial SAE section of the eCRFs, and provide any additional written documentation to the Safety Group immediately or within 1 working day of receipt.

The Sponsor or designee is responsible for notifying regulatory agencies of SAEs that require reporting as per the governing regulations.

It is the responsibility of the Investigator to report to the relevant IRB/EC in accordance with the IRB/EC's reporting specific reporting requirements for SAEs.

All SAEs must be followed up until the event is resolved, returns to the baseline condition, or is declared medically stable with no further change expected or the subject is lost to follow up.

**SAEs Occurring after the Follow-Up Visit**: If an SAE comes to the attention of the Investigator after study termination within 30 days of the last dose of study drug(s), and it is considered related to study drug, it must be recorded and followed up in the same way as the SAEs occurring during the study.

Any report of pregnancy identified for any female subject or for a female partner of a male subject should be reported immediately (within 24 hours of being informed) to the medical monitor. Pregnancies will be considered 'events of special interest' and will not be captured as serious adverse events (SAEs). The Pregnancy Report Form will be utilized to obtain follow-up information. Pregnancies will be followed to termination or eight weeks post-delivery for determination of resolution to the event. Subjects who become pregnant during the treatment period must immediately be withdrawn from the study (classified as ET). Subjects who become pregnant within 30 days following treatment must be reported to the sponsor.

### 8. STATISTICS

# 8.1. Sample Size Determination

A total of approximately 1400 subjects (approximately 700 in each treatment group) will be randomized.

For the co-primary endpoint of pain freedom at 2 hours post dosing of investigational drug, a therapeutic gain of 10%, assuming a 25% responder rate for STS101 and 15% for the placebo is targeted. Based on these assumptions, 700 subjects per arm can provide 99% power to detect the target treatment difference. For the co-primary endpoint of MBS freedom at 2 hours post investigational drug, a therapeutic gain of 10%, assuming a 45% responder rate for STS101 and 35% for the placebo is targeted. Based on these assumptions, 700 subjects per treatment group can provide 95% power to detect the target treatment difference. The sample size calculation is based on a chi-square test with a significance level of 0.05 and a 2-sided test.

The primary efficacy objective will be addressed by simultaneously testing the 2 co-primary endpoints of pain freedom and MBS freedom at 2 hours after drug administration at a significance level of 0.05. This sample size will provide an overall power of at least 94%.

### 8.2. Subject Populations

The analysis populations to be used in the study are defined below.

### **8.2.1** Intent-to-Treat Population

The intent-to-treat (ITT) population will include all randomized subjects who reported a qualifying migraine attack, received the study drug, and reported any post-treatment efficacy evaluation. Data will be analyzed according to the treatment group each subject is randomized to.

# 8.2.2 Modified Intent-to-Treat Population

For the purposes of efficacy data analysis, the modified intent-to-treat (mITT) population will be the primary analysis population. This population will include all randomized subjects who reported a qualifying migraine attack, received the study drug, and reported a post-treatment efficacy evaluation for at least 1 time point at or before the 2-hour time point. Data will be analyzed according to the treatment group each subject is randomized to.

# 8.2.3 Per-Protocol Population

The per protocol (PP) population will consist of all mITT subjects who do not have protocol deviations that could significantly affect the interpretation of the results for the primary endpoints. Subjects' inclusion/exclusion from the PP population will be determined and documented prior to the database lock and unblinding.

### 8.2.1. Safety Population

The safety population will include all subjects who are randomized and have received the study drug. Data will be analyzed according to the treatment each subject actually received.

# 8.3. Statistical Analysis

All study data will be summarized by treatment using descriptive statistics. Unless otherwise specified, for numeric data (e.g., age, weight), descriptive statistics will include the number of subjects with data to be summarized (n), mean, standard deviation (SD), median, minimum (min) and maximum (max). All categorical/qualitative data (e.g., gender, race) will be presented using absolute and relative frequency counts and percentage.

All summaries, statistical analyses, and individual subject data listings described below will be completed using Version 9.3 or later of the SAS software (SAS Institute, Inc. Cary, NC).

A detailed Statistical Analysis Plan (SAP) will be provided in a separate document. The SAP will include the final hierarchy for testing of the primary and secondary efficacy endpoints and will be finalized prior to database lock and unblinding of the study.

### 8.3.1. Demographic and Baseline Variables

Demographics and baseline characteristics (including migraine history, HIT-6 data and triptan response information) will be summarized descriptively by treatment group for the mITT Population, the ITT Population, the Per-Protocol Population, and the Safety Population. Exploratory hypotheses testing may be performed to assess the comparability of demographics and baseline characteristics among the treatment groups. No multiplicity adjustment will be applied to these tests.

### 8.3.2. Efficacy Analysis

### 8.3.2.1. Primary Efficacy Endpoints

- Proportion of subjects free from headache pain at 2 hours after dosing (defined as moderate or severe headache pain [2 or 3 on a 4-point scale] at baseline [time 0] becoming none [0] on a 4-point scale)
- Proportion of subjects free from most bothersome symptom (MBS) among photophobia, phonophobia and nausea at 2 hours after dosing (defined as the MBS identified at baseline [time 0] being absent)

### 8.3.2.2. Secondary Efficacy Endpoints

• Proportion of subjects with relief from headache pain at 2 hours after dosing (defined as reduction in headache pain from moderate or severe [2 or 3 on a 4-point scale] to mild or none [0 or 1 on a 4-point scale])

- Proportion of subjects who use rescue medication within 24 hours after dosing
- Proportion of subjects who achieve normal function at 2 hours after dosing (defined as score of 0 on the 4-point functional impairment scale)
- Proportion of subjects free from headache pain at 2 hours after dosing and remaining headache free at 24 hours after dosing with no use of rescue medication and no relapse of any headache pain (defined as score of 0 on a 4-point scale from 2-24 hours)
- Proportion of subjects free from headache pain at 2 hours after dosing and remaining headache free at 48 hours after dosing with no use of rescue medication and no relapse of any headache pain (defined as score of 0 on a 4-point scale from 2-48 hours)
- Proportion of subjects free from most bothersome symptom (MBS) at 2 hours after dosing and remaining MBS free at 24 hours after dosing with no use of rescue medication and no relapse of any MBS (defined as MBS selected at baseline [time 0] absent from 2-24 hours)
- Proportion of subjects free from most bothersome symptom (MBS) at 2 hours after dosing and remaining MBS free at 48 hours after dosing with no use of rescue medication and no relapse of any MBS (defined as MBS selected at baseline [time 0] absent from 2-48 hours)
- Proportion of subjects who use rescue medication within 48 hours after dosing
- Proportion of subjects with headache relapse within 24 hours after dosing (defined as the return of headache of any severity within 24 hours post dosing of the investigational drug, when the subject was pain-free at 2 hours after dosing)
- Proportion of subjects with headache relapse within 48 hours after dosing (defined as the return of headache of any severity within 48 hours post dosing of the investigational drug, when the subject was pain-free at 2 hours after dosing)
- Proportion of subjects free from headache pain at various time points after dosing
- Proportion of subjects free from most bothersome symptom at various time points after dosing
- Proportion of subjects achieving pain relief at various time points after dosing
- Proportion of subjects who achieve normal function at various timepoints after dosing
- Proportion of subjects free from photophobia at 2 hours after dosing (defined as photophobia being absent at 2 hours after dosing if present at baseline [time 0])
- Proportion of subjects free from phonophobia at 2 hours after dosing (defined as phonophobia being absent at 2 hours after dosing if present at baseline [time 0])
- Proportion of subjects free from nausea at 2 hours after dosing (defined as nausea being absent at 2 hours after dosing if present at baseline [time 0])
- Proportion of subjects free from photophobia at various timepoints after dosing
- Proportion of subjects free from phonophobia at various timepoints after dosing
- Proportion of subjects free from nausea at various timepoints after dosing
- Patient Global Impression ratings

### **8.3.2.3.** Exploratory Endpoints

• Proportion of subjects free from headache pain at 2 hours after dosing by allodynia status at baseline (allodynia status will be defined as "present" with at least 2 "yes" responses to the 6-question allodynia questionnaire [Ashkenazi 2007; Tepper 2011])

- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at 2 hours after dosing in subjects who wake up with migraine headache
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at 2 hours after dosing in subjects with menstrual related migraine attack
- Proportion of subjects with relief from headache pain at various timepoints after dosing by allodynia status at baseline (time 0) (allodynia status will be defined as "present" with at least 2 "yes" responses to the 6-question allodynia questionnaire [Ashkenazi 2007; Tepper 2011])
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at various timepoints after dosing in subjects who wake up with migraine headache
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at various timepoints after dosing in subjects with menstrual related migraine attack
- Proportion of subjects free from both, headache pain <u>and</u> most bothersome symptom (MBS) at 2 hours after dosing
- Proportion of subjects free from both, headache pain <u>and</u> most bothersome symptom (MBS) at various time points after dosing
- Proportion of subjects free from headache pain and free from most bothersome symptom (MBS) at 2 hours after dosing by baseline (Visit 2) HIT-6 score
- 24-hour Migraine Quality of Life Questionnaire summary scores

### 8.3.3. Hypotheses Testing and Significance Level

A study-wise Type I error of 0.05 will be used for this study. A multiplicity strategy will be taken into account when interpreting the nominal 2-sided p-values.

A fixed-sequence testing method which tests each endpoint individually in a pre-determined hierarchal order will be used for both primary and secondary endpoints. If the first endpoint is significant (<0.05), then you continue to the next endpoint. If an endpoint is not significant, then testing stops and all subsequent endpoints are considered non-significant.

The order of the secondary endpoints to be tested will be described in detail in the SAP.

# 8.3.4. Handling of Missing Data

For the primary analysis of the co-primary endpoints, missing data will be imputed based on a single-imputation method. Subjects who do not have evaluable assessments at the 2-hour time point, or who received rescue medications prior to the 2-hour time point will be considered as non-responders. The impact of missing data will be further investigated in a number of sensitivity analyses with other single and multiple-imputation approaches. The details of the sensitivity analyses will be described in the SAP.

### **8.3.5.** Pooling of Centers

Data from all investigational centers will be pooled for analysis. The analyses will not be performed by center and will not include adjustment for centers.

### 8.3.6. Analysis Methods for Efficacy Endpoints

For both co-primary endpoints, the Chi-square test will be used to compare the active treatment group and placebo. The Chi-square test will also be used to test the secondary endpoints defined as a response variable. For analyses stratified by allodynia status, timing of treatment, or any other baseline characteristic the Cochran-Mantel-Haenszel test will be used. The Kaplan-Meier method will be used for time to use of rescue medications. The 24-hour Migraine Quality of Life Questionnaire assessments will be analyzed with the Analysis of Variance (ANOVA) models. The Chi-Square test will be used to analyze the Patient Global Impression ratings.

To fully describe the treatment benefit of STS101, the proportion of subjects achieving "no headache pain" at various time points following treatment will be tested between the active treatment groups and placebo. The results will also be displayed graphically to show the time course of effect. To address the onset of efficacy, treatment difference vs. placebo will be examined from the 2 hour-timepoint towards the baseline in a sequential manner (i.e., 2 hours, 1.5 hours, 1 hour, 45 minutes, 30 minutes, 15 minutes). A significance level of 0.05 will be used for this analysis.

### 8.3.7. Subgroup Analysis of Efficacy Endpoints

Subgroup analyses of the key efficacy endpoints will be conducted to gain insight of the nature and consistency of the treatment effect. Subgroups prospectively identified include:

- 1. age group
- 2. gender
- 3. race
- 4. baseline severity of attack (time 0)
- 5. allodynia status
- 6. menstrual related migraine attacks
- 7. in subjects who wake up with migraine headache
- 8. baseline (Visit 2) HIT-6 score

Among these subgroup analyses, # 4, 5, 6, 7, and 8 are also included in the secondary or exploratory endpoints. Analysis by additional subgroups may be considered. They will be specified in the SAP before the study is unblinded for analysis.

Because of the smaller sample sizes for each subgroup, the objective of the analysis is to evaluate the consistency of efficacy results across these factors. Statistical tests will be performed. However, the interpretation of the p-values will take into account sample size and multiplicity issues. Forest plots with estimates and 95% confidence intervals of the treatment effect across different subgroups will be presented.

### 8.3.8. Safety Analysis

Safety analyses will be conducted for the safety population, which will include all subjects who received at least one dose of study medication. All clinical safety and tolerability data will be summarized by treatment group and listed by treatment group and by subject. All reported

adverse events will be coded using MedDRA and listed by System Organ Class, Preferred Term, and verbatim term. No inferential statistics will be performed; only summary statistics will be provided unless otherwise noted. Missing safety data will not be imputed.

### 8.3.8.1. Extent of Exposure

The number of subjects exposed to each treatment group will be summarized. Because this is a single-dose study, each subject is expected to receive one dose only.

### 8.3.8.2. Adverse Events

A TEAE is defined as an AE that begins after the dosing of study drug.

An overview of adverse events will be presented by treatment group, which will include the number and percent of subjects who had at least one AE, TEAE, Serious TEAE, TEAE related to study drug, and maximum severity of TEAE.

Multiple occurrences of an AE are counted only once per subject per SOC and PT for summary tables.

The following TEAEs will be summarized by SOC, PT and treatment group:

- Incidence of all TEAEs
- Nasal TEAEs (including taste sensations coded as dysgeusia)
- Incidence of all TEAEs by maximum severity (severe, moderate and mild) specified by investigators
- Incidence of TEAEs related to the study drug as determined by the investigators
- Incidence of serious TEAEs

All data collected in the AE case report form (CRF) will be listed in by-subject listings.

### **8.3.8.3.** Assessment of Nasal Symptoms

The data from the Objective Assessment of Nasal Symptoms (Appendix C) will be summarized by treatment group. Exploratory hypothesis testing may be performed to compare treatment group by question. No multiplicity adjustment will be applied to these tests.

### **8.3.8.4.** Laboratory Evaluations

The observed data at each time point and change from screening (Visit 1 or if re-draw: qualifying value) to the final study visit (Visit 3) in hematology, serum chemistry and quantitative urinallysis test results will be summarized by treatment group.

For hematology and serum chemistry including calculated creatinine clearance, normal ranges for each parameter will be used to categorize the test result as low (value lower than the lower limit), normal (value within the normal range), or high (value higher than the upper limit). For

urinalysis, test results will be categorized as normal and abnormal. Frequency counts and percentages will be presented over time by treatment groups for these categorical data. In addition, shifts from baseline (shift to maximum value, shift to minimum value) to each post-baseline time point and to any post-baseline time point for each parameter will be summarized by treatment group.

If a continuous laboratory value is reported as either below or above the limits of quantification, the qualifiers should be dropped and the numeric value used in the analysis (e.g., "< 1" should be "1" and "> 100" should be "100").

### **8.3.8.5.** Vital Signs

Observed data at each time point and the change from baseline (Visit 2) at each post-baseline time point for vital signs will be summarized by treatment group.

Normal ranges for each vital sign parameter will be used to categorize the results as low (lower than the lower limit), normal (within the normal range), or high (higher than the upper limit). Frequency counts and percentages will be presented over time by treatment group for these categorical data.

### **8.3.8.6.** ECG Evaluations

Observed data at each time point and the change at baseline (Visit 2) at each post-baseline time point in ECG parameters, heart rate (HR), RR, PR, QRS, and QT corrected with the Fridericia's formula (QTcF), will be summarized by treatment groups.

The number and percentage of subjects with other clinically significant ECG findings will also be summarized at each post baseline time point by treatment group.

#### **8.3.8.7.** Concomitant Medications

Concomitant medication usage will be summarized by the number and proportion of subjects in each treatment group. The World Health Organization Drug Dictionary (WHO Drug) will be used to classify prior and concomitant medications by therapeutic class and generic name based on ATC code level 3. Subjects will only be counted one time in each unique ATC Class and generic name if multiple drugs are used by a subject.

### 8.3.8.8. Sheehan Suicidality Tracking Scale

Reported data at each time point and the change from baseline (Visit 1) at Visit 3 will be summarized by treatment groups.

### 8.3.9. Interim analysis

No interim analysis is planned for this study.

### 9. DATA HANDLING AND RECORDKEEPING

# 9.1. Case Report Forms (CRFs)

All clinical study data will be collected by the clinical investigator and staff, recorded on source documents and captured electronically in the electronic CRF.

The populated electronic CRFs will be monitored against source documents by the Sponsor's representative and any subsequent data discrepancies identified will be recorded and communicated to the investigative site for resolution.

Completion of the electronic CRF should occur within 24 hours of a subject's visit.

## 9.2. Retention of Records

The Investigator must maintain adequate records for the study including all source documentation, completed CRFs, logs, medical records, laboratory reports, signed ICFs, investigational product disposition records, adverse event reports, information regarding subjects who discontinued, all correspondence with the EC and the Sponsor (or designee) and other pertinent data.

The study site will maintain adequate study records for at least 2 years after product approval for marketing or until instructed by the Sponsor in writing. After that period, the Sponsor may be contacted to determine whether the study records will be forwarded to the Sponsor, destroyed or kept at another facility for a longer period of time at the Sponsor's expense.

To avoid any possible errors, the Investigator must contact Satsuma (or designee) prior to the destruction of any study records. The Investigator will also notify Satsuma (or designee) in the event of accidental loss or destruction of any study records.

# 10. QUALITY CONTROL AND QUALITY ASSURANCE

# 10.1. Study Monitoring

The study will be monitored by the Sponsor's representatives at all stages of study conduct from inception to completion in accordance with current Good Clinical Practice (GCP) guidelines. This monitoring will be in the form of site visits and other communication and will include review of original source documents and CRFs. The Sponsor's monitor or representative will notify the Principal Investigator prior to conducting any investigational site visit. The frequency of these visits will depend upon the progress of the study, and will include monitoring to assess facilities and equipment, recruiting, record-keeping, protocol adherence, data collection, investigational product accountability, AE reporting and other factors.

# 10.2. Audits and Inspections

The clinical site will be subject to audit and inspection by the Sponsor or representative during and/or at the end of the study as appropriate.

The Investigator will permit representatives of Satsuma or representative or FDA auditors to inspect facilities and records relevant to this study, including the subject's original medical records for verification of study-related procedures and data.

### 11. ETHICS

### 11.1. Ethics Review

The Ethics Committee/Institutional Review Board will review and approve the study protocol, the ICF and other relevant substantive information or documents before the study is initiated. If an Investigator chooses to advertise for subjects for this study, whether in professional or consumer publications, radio, or television or any digital media, all advertising copy and language must be approved by Satsuma and the EC/IRBs prior to initiation.

A copy of the EC/IRB approval letter for the protocol and the consent form/subject information sheet, which specifically identifies the protocol name and the Satsuma protocol number, must be sent to Satsuma (or designee) prior to initiating the study. Subsequently, the Investigator is responsible for keeping the EC/IRB advised of the progress of the study as deemed appropriate but, in any case, at least once a year during the course of the study and for keeping the EC/IRB informed of any significant study change or adverse reactions per EC/IRB specific guidelines.

# 11.2. Ethical Conduct of the Study

This study will be conducted in strict compliance with the Declaration of Helsinki, ICH, GCP, EC/IRB and other relevant regulatory requirements and laws.

The Investigator must ensure that each subject's anonymity is maintained as described within this protocol. On the CRFs or other documents submitted to Satsuma, or its designee, subjects must be identified only by their initials and a subject number. Documents that are not for submission to Satsuma, and/or its designee, (i.e., signed ICFs) should be kept in strict confidence by the Investigator, in compliance with Federal regulations and ICH and GCP Guidelines. The Investigator is obligated to inform the subject in the ICF that his/her study-related records will be reviewed by the above-named study sponsor and representatives.

### 11.3. Written Informed Consent

Prior to any study procedures being performed, each study participant will be required to read, sign and date an EC/IRB -approved ICF, explaining the nature, purpose, possible risks and benefits, and the duration of the study.

The ICF must be written in English or Spanish, and all subjects must be fluent in English or Spanish (speaking, writing, and reading). The Investigator or designee shall give the subject, adequate time to read the ICF and consider study participation and have all questions answered. They should also express understanding of the information presented regarding the trial before it is signed and dated.

The ICF must contain the subject's dated signature confirming the consent. In addition, a witness must also sign and date the ICF. The person who conducted the informed consent discussion will

also be sign and date the consent form. Each participant will be given a copy of the fully executed ICF.

Each subject's signed ICF must be kept on file by the Investigator and be available for possible inspection by regulatory authorities, and/or the study Sponsor or designee, or the EC/IRB. Documentation of the informed consent and subject information discussion must appear in the subject's medical record and/or the subject's study file and be available for verification by monitors at any time.

### 11.4. Disclosure of Data

Individual subject medical information obtained as a result of this study is considered confidential, and disclosure to third parties other than those noted below is prohibited.

However, at the request of the subject such medical information may be given to the subject's personal physician, or to other appropriate medical personnel responsible for the subject's welfare.

In addition, data generated during this study are to be available for inspection upon request by FDA auditors, the Sponsor's monitors or by the EC/IRB. Therefore, absolute confidentiality cannot be guaranteed.

The sponsor is planning a publication of the complete study data. No publication of an individual site's data may occur before that publication and no publications may occur without the sponsor's written approval.

### 12. REFERENCES

Ashkenazi A, Sholtzow M, Shaw JW, Burstein R, Young WB. Identifying cutaneous allodynia in chronic migraine using a practical clinical method. Cephalalgia. 2007;27(2):111-7. doi: 10.1111/j.1468-2982.2006.01255.x.

Aurora SK, Silberstein SD, Kori SH, Tepper SJ, Borland SW, Wang M, Dodick DW. MAP0004, orally inhaled DHE: a randomized, controlled study in the acute treatment of migraine. Headache. 2011;51(4):507-17. doi: 10.1111/j.1526-4610.2011.01869.x.

Burstein R, Collins B, Jakubowski M. Defeating migraine pain with triptans: a race against the development of cutaneous allodynia. Ann Neurol. 2004;55(1):19-26. doi: 10.1002/ana.10786.

Carleton SC, Shesser RF, Pietrzak MP, Chudnofsky CR, Starkman S, Morris DL, Johnson G, Rhee KJ, Barton CW, Chelly JE, Rosenberg J, Van Valen MK. Double-blind, multicenter trial to compare the efficacy of intramuscular dihydroergotamine plus hydroxyzine versus intramuscular meperidine plus hydroxyzine for the emergency department treatment of acute migraine headache. Ann Emerg Med. 1998;32(2):129-38.

Cook RO, Shrewsbury SB, Ramadan NM. Reduced adverse event profile of orally inhaled DHE (MAP0004) vs IV DHE: potential mechanism. Headache. 2009;49(10):1423-34. doi: 10.1111/j.1526-4610.2009.01510.x.

D.H.E. 45® Prescribing Information. Bridgewater (NJ): Valeant Pharmaceuticals; 2017 Nov.

Dahlöf C, Maassen Van Den Brink A. Dihydroergotamine, ergotamine, methysergide and sumatriptan - basic science in relation to migraine treatment. Headache. 2012;52(4):707-14. doi: 10.1111/j.1526-4610.2012.02124.x.

Diener H-C, Ferrari M, Mansbach H. Predicting the response to sumatriptan: the Sumatriptan Naratriptan Aggregate Patient Database. Neurology. 2004;63(3):520-4. doi: 10.1212/01.wnl.0000133207.70312.30.

Diener H-C, Tassorelli C, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ, Mandrekar J, International Headache Society Clinical Trials Standing C. Guidelines of the International Headache Society for controlled trials of acute treatment of migraine attacks in adults: Fourth edition. Cephalalgia. 2019:333102419828967. doi: 10.1177/0333102419828967.

Djupesland PG, Messina JC, Mahmoud RA. Breath powered nasal delivery: a new route to rapid headache relief. Headache. 2013;53 Suppl 2:72-84. doi: 10.1111/head.12186.

Dodick DW, Lipton RB, Ailani J, Lu K, Finnegan M, Trugman JM, Szegedi A. Ubrogepant for the Treatment of Migraine. New England Journal of Medicine. 2019;381(23):2230-41. doi: 10.1056/NEJMoa1813049.

Edwards KR, Norton J, Behnke M. Comparison of intravenous valproate versus intramuscular dihydroergotamine and metoclopramide for acute treatment of migraine headache. Headache. 2001;41(10):976-80.

Gallagher RM. Acute treatment of migraine with dihydroergotamine nasal spray. Dihydroergotamine Working Group. Arch Neurol. 1996;53(12):1285-91.

Goadsby PJ, Wietecha LA, Dennehy EB, Kuca B, Case MG, Aurora SK, Gaul C. Phase 3 randomized, placebo-controlled, double-blind study of lasmiditan for acute treatment of migraine. Brain. 2019;142(7):1894-904. doi: 10.1093/brain/awz134.

González-Hernández A, Lozano-Cuenca J, Marichal-Cancino BA, MaassenVanDenBrink A, Villalón CM. Dihydroergotamine inhibits the vasodepressor sensory CGRPergic outflow by prejunctional activation of α2-adrenoceptors and 5-HT1 receptors. The Journal of Headache and Pain. 2018;19(1):40. doi: 10.1186/s10194-018-0869-8.

Hartmaier SL, Santanello NC, Epstein RS, Silberstein SD. Development of a brief 24-hour migraine-specific quality of life questionnaire. Headache. 1995;35(6):320-9.

Hoskin KL, Kaube H, Goadsby PJ. Central activation of the trigeminovascular pathway in the cat is inhibited by dihydroergotamine. A c-Fos and electrophysiological study. Brain. 1996;119 (Pt 1):249-56.

Kuca B, Silberstein SD, Wietecha L, Berg PH, Dozier G, Lipton RB. Lasmiditan is an effective acute treatment for migraine: A phase 3 randomized study. Neurology. 2018;91(24):e2222-e32. doi: 10.1212/wnl.000000000006641.

Lipton RB, Dodick DW, Ailani J, Lu K, Finnegan M, Szegedi A, Trugman JM. Effect of Ubrogepant vs Placebo on Pain and the Most Bothersome Associated Symptom in the Acute Treatment of Migraine: The ACHIEVE II Randomized Clinical Trial. JAMA. 2019;322(19):1887-98. doi: 10.1001/jama.2019.16711.

Marmura MJ, Silberstein SD, Schwedt TJ. The acute treatment of migraine in adults: the american headache society evidence assessment of migraine pharmacotherapies. Headache. 2015;55(1):3-20. doi: 10.1111/head.12499.

Migranal® Administration Instructions. Valeant Pharmaceuticals.

Migranal® Prescribing Information. Aliso Viejo (CA): Valeant Pharmaceuticals.

Raskin NH. Repetitive intravenous dihydroergotamine as therapy for intractable migraine. Neurology. 1986;36(7):995-7.

Silberstein SD, McCrory DC. Ergotamine and dihydroergotamine: history, pharmacology, and efficacy. Headache. 2003;43(2):144-66.

Tepper SJ, Kori SH, Goadsby PJ, Winner PK, Wang MH, Silberstein SD, Cutrer FM. MAP0004, orally inhaled dihydroergotamine for acute treatment of migraine: efficacy of early and late treatments. Mayo Clin Proc. 2011;86(10):948-55. doi: 10.4065/mcp.2011.0093.

Tfelt-Hansen PC. Relatively slow and long-lasting antimigraine effect of dihydroergotamine is most likely due to basic pharmacological attributes of the drug: a review. Cephalalgia. 2013;33(13):1122-31. doi: 10.1177/0333102413483372.

van der Kuy PH, Lohman JJ, Hooymans PM, Ter Berg JW, Merkus FW. Bioavailability of intranasal formulations of dihydroergotamine. Eur J Clin Pharmacol. 1999;55(9):677-80.

Winner P, Ricalde O, Le Force B, Saper J, Margul B. A double-blind study of subcutaneous dihydroergotamine vs subcutaneous sumatriptan in the treatment of acute migraine. Arch Neurol. 1996;53(2):180-4.

Yang M, Rendas-Baum R, Varon SF, Kosinski M. Validation of the Headache Impact Test (HIT-6) across episodic and chronic migraine. Cephalalgia. 2010;31(3):357-67. doi: 10.1177/0333102410379890.

# Appendix A. Schedule of Assessments

| | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| | Screening | Randomization | Follow-up / Early Termination |
| Timing of Visit | Day -30 to -1 | Day 1 | Within one week (±3 days) of use of study medication<br>(no later than Study Day 66) |
| Informed consent | X | | |
| Demographic data / Medical history | X | | |
| Physical examination | X | X | X |
| Vital signs | X | X | X |
| Body weight and height | X | Xa | X <sup>a</sup> |
| BMI Calculation | X | | |
| Hematology, clinical chemistry, urinalysis <sup>f</sup> | X | | X |
| Serum & Urine pregnancy screen (All females) | Xg | X | Xg |
| Urine Drug and Alcohol Screen | X | | |
| 12-lead ECG (in triplicate) | X | | X |
| Determine / review eligibility | X | X | |
| HIT-6 Instrument | | X | |
| Sheehan Suicidality Tracking Scale (S-STS) | X | X | X |
| Headache Diary use training & review | X | X | X <sup>d</sup> |
| Headache Diary event recording | Xb | X <sup>c</sup> | |
| Objective Assessment of Nasal Symptom | X | X | X |
| Placebo Response Reduction Training | X | X | |
| Patient Subjective Impression Questions (6.2) | | | X |
| Randomization | | X | |
| Concomitant medications | X | X | X |
| STS101 Administration Training | X | X | |
| Investigational Product supply | | X | Xe |
| Adverse events recording | X | X | X |

<sup>&</sup>lt;sup>a</sup> Weight only; <sup>b</sup> Recording of headaches for 15 days; <sup>c</sup> Recording of headache severity & symptoms of treated attack, <sup>d</sup> Collect e-diary device; <sup>e</sup> Collect STS101 device; <sup>f</sup> FSH in menopausal females (surgical or physiologically menopausal); <sup>g</sup> Serum only

# Appendix B. List of Allowed and Disallowed Other Headache Types

Note: Subjects may not have 15 or more headache days per month in the three months before screening (Visit 1)

# a) Allowed headache types

Subjects may be included in the study if they have these types of headaches and if they can distinguish them from their migraines:

- Tension headache
- "Regular" headache
- Sinus congestion related headache
- Headache related to temporomandibular joint dysfunction
- Temporary headaches, e.g., from spinal tap or dental conditions that are temporary and no longer present when subject starts treatment period

Note: Subjects must be instructed not to treat any of the above listed headaches with study medication

### b) Disallowed headache types

- Medication overuse headache ("Regular intake of ergotamine or triptan on ≥10 days/month for >3 months")
- Post traumatic headache, e.g., within post-concussion syndrome
- Headache related to intracranial structures, e.g., intracranial neoplasm, aneurysm
- Headache related to other conditions, e.g., subarachnoid hemorrhage, acute or chronic subdural hematoma, intracranial infections or meningitis
- Basilar migraine, now called: "Migraine with Brainstem Aura" (MBA)
- Hemiplegic migraine
- Cluster headache
- Trigeminal neuralgia, other cranial neuralgias
- Temporal arteritis
- Intracranial inflammatory conditions or autoimmune related headaches.
- Chronic dental conditions that lead to headaches
- Intracranial hypertension (pseudotumor cerebri)
- Spinal headache (e.g., due to intracranial hypotension due to a CSF leak)

# Appendix C. Objective Assessment of Nasal Symptoms

A total of 5 questions are listed in this assessment sheet. On the numerical rating scale below, identify the degree of the presence of the **BOLD** physical finding by choosing a number from 0: none, 1: mild, 2: moderate, 3: severe. This sheet will be completed by the qualified physician or physician assistant or nurse practitioner who performs the examination.

### 1. Nasal Erythema (please circle)

| 0 | 1 | 2 | 3 |
|--------|--------|------------|----------|
| (none) | (mild) | (moderate) | (severe) |

Mild = redness limited to < 20 % of visible nasal mucosa

Moderate = redness 20-50 % of visible nasal mucosa Severe = redness > 50 % of visible nasal mucosa

### 2. Nasal Edema (please circle)

| | 0 | 1 | 2 | 3 |
|----|-------|--------|------------|----------|
| (r | none) | (mild) | (moderate) | (severe) |

Mild = localized swelling < 20 % of visible nasal mucosa Moderate = area of swelling 20-50 % of visible nasal mucosa Severe = swelling affects > 50 % of visible nasal mucosa

# 3. **Rhinorrhea** (please circle)\*

| 0 | 1 | 2 | 3 |
|--------|--------|------------|----------|
| (none) | (mild) | (moderate) | (severe) |

Mild = subject reports blowing nose < 3 times in 1 hour Moderate = subject reports blowing nose 4-7 times in 1 hour

Severe = subject reports blowing nose 8 or greater number of times in 1 hour

(continued on next page)

# 4. Nasal Bleeding (please circle)

| 0 | 1 | 2 | 3 |
|--------|--------|------------|----------|
| (none) | (mild) | (moderate) | (severe) |

Mild = blood streaking on tissue

Moderate = less than 5 mL (1 teaspoon) estimated bleeding

Severe = greater than or equal to 5 mL (1 teaspoon) estimated bleeding

# 5. Nasal Ulceration (please circle)



Mild = mucosal erosion < 2 mm in diameter Moderate = mucosal erosion 3-5 mm in diameter

Severe = mucosal erosion/ulceration 6 mm or greater in diameter

Signature of Investigator Date (dd/mm/yyyy)

# Appendix D. STS101 Instructions for Use



# Appendix E. 24-Hour Migraine Quality of Life Questionnaire

#### 24-HOUR MIGRAINE QUALITY OF LIFE QUESTIONNAIRE Only the patient (subject) should enter information onto this questionnaire. The following questions are to be completed 24 HOURS after you take your first dose of medication for your migraine headache, and ask how your quality of life was affected. In the past 24 HOURS after you took your first dose of medication for your migraine headache, how much of the time did you: (Please check one box for each question) All Most A good Some A little Hardly None of the of the bit of the of the of the any of the of the time time time time time time time 1 5 6 2 3 4 7 1. have increased sensitivity to light and/or noise ..... 2. have nausea ..... 3. have throbbing head pain ...... 4. feel upset about having migraine headaches ..... 5. feel physically uncomfortable ....... 6. feel concerned that your migraine medication wouldn't relieve your migraine headache symptoms ......

Copyright © 1995 Merck & Co., Inc. Whitehouse Station, N.J., U.S.A. All Rights Reserved

| 24-HOUR MIGRAIN | E QU | ALITY | OF LI | FE QU | ESTIC | NNAIR | E |
|---|---|---|---|---|---|---|---|
| In the past 24 HOURS after you took your first dose of medication, how much of the time did your migraine headache and accompanying symptoms limit your ability to: (Please check <u>one</u> box for each question) | | | | | | | |
| | All<br>of the<br>time<br>1 | Most of the time | A good<br>bit of the<br>time<br>3 | Some<br>of the<br>time | A little of the time | Hardly<br>any of the<br>time<br>6 | None<br>of the<br>time<br>7 |
| 7. do normal everyday work (job outside the home, schoolwork, housework) | 🗆 | | | | | | |
| 8. stay alert | | | | | | | |
| operate machinery or a motor<br>vehicle (including home appliance<br>and office equipment) | | | | | | | |
| 10. enjoy life | 🗌 | | | | | | |
| In the past 24 HOURS after you took your first dose of medication, how much did your migraine headache and accompanying symptoms <u>negatively</u> affect your: | | | | | | | |
| | nd acco | mpanyin | | | | | |
| your migraine headache ai | A very great deal | mpanyin<br>stion)<br>A great<br>deal | g sympte<br>A good<br>deal | A<br>moderate<br>amount | Some | Very | :<br>None |
| your migraine headache and (Please check one box for expectation) | nd accor<br>ach ques<br>A very<br>great | mpanyin<br>stion)<br>A great | <b>g sympt</b> o | A<br>moderate | atively a | ffect your | : |
| your migraine headache ai | A very great deal | mpanyin<br>stion)<br>A great<br>deal | g sympte<br>A good<br>deal | A<br>moderate<br>amount | Some | Very | :<br>None |
| your migraine headache au (Please check <u>one</u> box for el 11. interactions with people who | A very great deal 1 | mpanyin<br>stion)<br>A great<br>deal | g sympte<br>A good<br>deal | A<br>moderate<br>amount | Some | Very | :<br>None |
| your migraine headache au (Please check one box for el 11. interactions with people who are close to you | A very great deal 1 | mpanyin<br>stion)<br>A great<br>deal | g sympte<br>A good<br>deal | A<br>moderate<br>amount | Some | Very | :<br>None |
| your migraine headache au (Please check one box for el 11. interactions with people who are close to you | A very great deal 1 | mpanyin<br>stion)<br>A great<br>deal | g sympte<br>A good<br>deal | A<br>moderate<br>amount | Some | Very | :<br>None |
| your migraine headache au (Please check one box for extended one) 11. interactions with people who are close to you | A very great deal 1 | mpanyin<br>stion)<br>A great<br>deal | g sympte<br>A good<br>deal | A<br>moderate<br>amount | Some | Very | :<br>None |

Copyright © 1995 Merck & Co., Inc. Whitehouse Station, N.J., U.S.A. All Rights Reserved

Reference: Hartmaier 1995

# Appendix F. Headache Impact Test (HIT-6<sup>TM</sup>)

# HIT-6<sup>TM</sup>

# HEADACHE IMPACT TEST

This questionnaire was designed to help you describe and communicate the way you feel and what you cannot do because of headaches.

To complete, please check one box for each question.

| 1. \ | When you have hea | adaches, how ofte | en is the pain severe? | | |
|---|---|---|---|---|---|
| | ☐ Never | Rarely | ☐ Sometimes | ☐ Very Often | ☐ Always |
| | How often do head<br>work, work, school | _ | bility to do usual daily<br>es? | activities including | household |
| | □ Never | Rarely | ☐ Sometimes | ☐ Very Often | ☐ Always |
| 3. ۱ | _ | | en do you wish you co | | |
| | □ Never | Rarely | ☐ Sometimes | ☐ Very Often | ☐ Always |
| | n the past 4 weeks<br>your headaches? | , how often have | you felt too tired to do | work or daily activi | ties because of |
| | ■ Never | Rarely | ☐ Sometimes | ☐ Very Often | ☐ Always |
| 5. ı | n the past 4 weeks | s, how often have | you felt fed up or irrita | ted because of you | headaches? |
| | □ Never | ☐ Rarely | ☐ Sometimes | ☐ Very Often | ☐ Always |
| | n the past 4 weeks<br>activities? | s, how often did he | eadaches limit your ab | ility to concentrate | on work or daily |
| | ■ Never | ☐ Rarely | ☐ Sometimes | ☐ Very Often | ☐ Always |

# **Appendix G.** Sheehan Suicidality Tracking Scale (S-STS)

# SHEEHAN-SUICIDALITY TRACKING SCALE (S-STS)

INSTRUCTIONS: PLEASE USE DATA FROM ALL SOURCES AND CONSIDER SEVERITY, FREQUENCY, TIME SPENT AND TIME FRAME IN YOUR RESPONSES. THE RESPONSE
"NOT AT ALL" TO ANY QUESTION MEANS "NONE" AND MEANS THAT THE THOUGHT, EXPERIENCE OR BEHAVIOR "DID NOT OCCUR AT ALL". THROUGHOUT THE
SCALE, THE WORDS INTENT / INTEND MEAN ANY INTENT GREATER THAN ZERO. SCORE THE MOST SERIOUS EVENT THAT OCCURRED FOR EACH ITEM BELOW.

| In t | he past (timeframe): | | | | | |
|---|---|---|---|---|---|---|
| 1. | did you have any accident? (this includes taking too much of your medication accidentally) IF NO, SKIP TO QUESTION 2. IF YES, GO TO QUESTION 1a: | | NO | | YES [ | ] |
| 12. | how seriously did you plan or intend to hurt yourself in any accident, either by not avoiding a risk or by causing the accident on purpose? IF THE ANSWER TO QUESTION 1a IS 0 (= Not at all), SKIP TO QUESTION 2. IF THE SCORE IS 1 OR HIGHER, GO TO QUESTION 1b: | Not at all | A little | Moderately 2 | Very<br>3 | Extremely 4 |
| 1b. | did you intend to die as a result of any accident? | | NO I | | YES [ | |
| In t | he past (timeframe), how seriously did you:<br>think (even momentarily) that you would be better off dead, need to be dead<br>or wish you were dead?<br>How many times? | Not at all | A little | Moderately 2 | Very<br>3 | Extremely 4 |
| 3. | think (even momentarily) about harming or hurting or injuring yourself — with at least some intent or awareness that you might die as a result — or think about suicide (killing yourself)? How many times? | 0 | 1 | 2 | 3 | 4 |
| 4. | have a voice or voices telling you to kill yourself or have dreams with any suicidal content? mark either or both; a voice or voices a dream | 0 | 1 | 2 | 3 | 4 |
| 5. | have any suicide method in mind (i.e. how)? # | 0 | 1 | 2 | 3 | 4 |
| 6. | have any suicide means in mind (i.e. with what)?# | 0 | 1 | 2 | 3 | 4 |
| 7. | have any place in mind to attempt suicide (i.e. where)? * # | 0 | 1 | 2 | 3 | 4 |
| 8. | have any date / timeframe in mind to attempt suicide (i.e. when)?*# | 0 | 1 | 2 | 3 | 4 |
| 9. | intend to act on thoughts of killing yourself?<br>mark either or both: did you intend to act: $\square$ at the time $\square$ at some time in the future | 0 | 1 | 2 | 3 | 4 |
| 10. | intend to die as a result of a suicidal act? mark either or both: did you intend to die: at the time at some time in the future | 0 | 1 | 2 | 3 | 4 |
| 11. | feel the need or impulse to kill yourself or to plan to kill yourself sooner rather than later? mark either or both: was this: | 0 | 1 | 2 | 3 | 4 |
| 12. | take active steps to prepare for a suicide attempt in which you expected or intended to die (include anything done or purposely not done that put you closer to making a suicide attempt)? | 0 | 1 | 2 | 3 | 4 |
| 13. | injure yourself on purpose without intending to kill yourself? How many times? | 0 | 1 | 2 | 3 | 4 |
| 14. | attempt suicide (try to kill yourself)? | 0 | 1 | 2 | 3 | 4 |

"A suicide attempt is a potentially self-injurious behavior, associated with at least same intent (> 0) to die as a result of the act. Evidence that the individual intended to kill him- or herself, at least to same degree, can be explicit or inferred from the behavior or circumstance.

A suicide attempt may or may not result in actual injury." (FDA 2012 definition 1.2). \* Note: Items 7 & 8 on S-STS ("a plan for suicide") means not going beyond ideas or talking about a plan for suicide. If actual behaviors occurred, the event should not be coded on item 7 or 8, but as "preparatory behavior" (item 12). Both events can occur separately over the same timeframe. # Note: clinician should ask for details.

# SHEEHAN-SUICIDALITY TRACKING SCALE (S-STS) - EVENTS REPORT

| Not at all | | | | | |
|---|---|---|---|---|---|
| | A little | Moderately | Very | Extremely | Level |
| 0 | 1 | 2 | 3 | 4 | 3 |
| 0 | 1 | 2 | 3 | 4 | |
| 0 | 1 | 2 | 3 | 4 | |
| 0 | 1 | 2 | 3 | 4 | |
| 0 | 1 | 2 | 3 | 4 | 7 |
| e interrupted a<br>as you meant to | | t finish the | attemp | t. | |
| e interrupted a<br>as you meant to | | t fin <mark>i</mark> sh the | attemp | t. | |
| e steps to prep<br>done that put | o.<br>oare for a<br>you close | suicide atte<br>r to making | empt in | which you | |
| e steps to <u>prep</u><br>done that put v | o.<br><u>pare</u> for a<br>you close<br>le attemp | suicide atte<br>r to making | empt in<br>a suicid | which you<br>de attempt | |
| e steps to <u>prep</u><br>done that put v | o.<br><u>pare</u> for a<br>you close<br>le attemp | suicide atte<br>r to making<br>pt.) | empt in<br>a suicid<br>aration? | which you<br>de attempt | |
| e steps to <u>prep</u><br>done that put y<br>an actual suicid | o.<br>pare for a<br>you close<br>le attemp<br>rious was | suicide atte<br>r to making<br>ot.)<br>s each prepa | empt in<br>a suicid | which you<br>de attempt | :)? |
| e steps to <u>prep</u><br>done that put y<br>an actual suicid<br>How se | o.<br>oare for a<br>you close<br>le attemp<br>rious was | suicide atte<br>r to making<br>ot.)<br>s each prepa<br>Moderately | empt in<br>a suicid<br>aration?<br>Very | which you<br>de attempt | :)? |
| e steps to prep<br>done that put<br>an actual suicid<br>How se | o. oare for a you close le attemprious was | suicide atte<br>r to making<br>st.)<br>each prepa<br>Moderately | empt in a suicid | which you le attempt | :)? |
| e steps to prepdone that put the an actual suicide How se | o. oare for a you close le attemprious was: | suicide atter to making st.) seach prepa | empt in a suicideration? | which you de attempt | :)? |
| | 0 0 0 nt, or not at all | 0 1 0 1 0 1 nt, or not at all) | 0 1 2 | 0 1 2 3<br>0 1 2 3<br>0 1 2 3 | 0 1 2 3 4 0 1 2 3 4 0 1 2 3 4 1 0 1 2 3 4 |

TIME SPENT PER DAY WITH ANY SUICIDAL IMPULSES, THOUGHTS OR ACTIONS OVER THE PAST (TIMEFRAME):

Level 3: You were about to try to kill yourself, but then someone or something stopped you just before harming yourself.

Usual time spent per day: hours minutes.

Least amount of time spent in any day: hours minutes.

Most amount of time spent in any day: hours minutes.

1/9/19

© Copyright Sheehan DV 2005-2019. All rights reserved. Permissions:davidvsheehan@gmail.com

FOR CLINICIAN USE ONLY

### SHEEHAN-SUICIDALITY TRACKING SCALE (S-STS) - CLINICIAN USE ONLY

Complete this section only if the patient does not return for the scheduled follow up visit and is not available to permit completion of pages 1 and 2. Only one response can be selected from 17 through 22.

| 17. N | lissed appointm | ent - reason: subject died fro | n a completed suicide? | | NO<br>0 | YES<br>100 |
|---|---|---|---|---|---|---|
| 18. N | lissed appointm | ent - reason: subject died, bu | t not enough information to code as a suicide | 7 | 0 | ** |
| 19. N | lissed appointm | ent - reason: subject died fro | n cause(s) other than suicide? | | 0 | ** |
| 20. N | lissed appointm | ent - reason: subject alive, bu | t not available because of a suicide attempt? | | 0 | 56 |
| 21. N | lissed appointm | ent - reason: subject alive, bu | t not available for known reasons other than | suicide? | 0 | ** |
| 22. N | lissed appointm | ent - reason: subject alive, bu | t not available, for uncertain reasons, or "lost | t to follow up"? | 0 | ** |
| Tot | al Scale Score | [the highest of 12 or any ro<br>15] or (only if applicable 17 | 1a (only if 1b is coded YES), + 2 through 11 + w of 16] + [the highest of 14 or any row of or 18 or 19 or 20 or 21 or 22 [page 3]). ** = prior visit only if this response is applicable. | TOTAL | | |
| | I have reviewed | I the answers on Pages 1 and | 2 with the patient. | | | |
| | Clinician Signat | ıre | dd/MMM/yyyy | | | |
| | I have reviewed | the answers on Pages 1 and | 2 with my doctor or clinician. | | | |
| | Patient Signatu | re | dd/MMM/yyyy | | | |

#### References

- Posner K, Oquendo MA et al. Columbia Classification Algorithm of Suicide Assessment (C-CASA): Classification of Suicidal Events in the FDA's Pediatric Suicidal Risk Analysis of Antidepressants. C-CASA Definitions in Table 2, page 1037. Am J Psychiatry 2007; 164:1035-1043

The author is grateful to JM Giddens for very valuable advice in the development of the S-STS and of the S-STS CMCM versions.

1/9/19